A Randomized, Double-blind, Placebo-controlled, Parallel-group,

Official Title: Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Added to a Sulfonylurea alone or in combination with Metformin in Patients with Type 2 Diabetes Who Have Inadequate

Glycemic Control on a Sulfonylurea Alone or with Metformin

NCT Number: NCT03066830

**Document Date(s):** SAP Version 3: 20 February 2020

# Lexicon Pharmaceuticals, Inc.

Protocol No.: EFC14835

A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Sotagliflozin Added to a Sulfonylurea alone or in combination with Metformin in Patients with Type 2 Diabetes Who Have Inadequate Glycemic Control on a Sulfonylurea Alone or with Metformin

Covance Study ID: 000000154257

# **Statistical Analysis Plan**

Version: 3

DATE OF ISSUE: 19 February 2020

Author:

#### APPROVALS

Printed Name/Title

The undersigned agree that all required reviews of this document are complete, and approve this Statistical Analysis Plan as final. Programming of the tables, figures and listings based upon the specifications within this document can proceed.

# **VERSION HISTORY**

| Version Status | Version Date |
|----------------|------------------|
| Final 1.0 | 07 August 2018 |
| Final 2.0 | 03 June 2019 |
| Final 3.0 | 19 February 2020 |

#### **TABLE OF CONTENTS**

| Α | PF | <u>'R</u> | <u>٥٧</u> | /A | <u>LS</u> |
|---|----|-----------|-----------|----|-----------|

## **VERSION HISTORY**

### **TABLE OF CONTENTS**

### **LIST OF ABBREVIATIONS AND DEFINITION OF TERMS**

| 1 0\ | /ERVIEW | AND INV | /ESTIGAT | IONAL | PLAN |
|------|---------|---------|----------|-------|------|

- 1.1 STUDY DESIGN AND RANDOMIZATION
- 1.2 OBJECTIVES
- 1.2.1 Primary objectives
- 1.2.2 Secondary objectives
- 1.2.3 Other objectives
- 1.3 DETERMINATION OF SAMPLE SIZE
- 1.4 STUDY PLAN
- 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL
- 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

#### 2 STATISTICAL AND ANALYTICAL PROCEDURES

- 2.1 ANALYSIS ENDPOINTS
- 2.1.1 Demographic and baseline characteristics
- 2.1.2 Prior or concomitant medications
- 2.1.2.1 Rescue therapy
- 2.1.2.2 Prohibited prior and concomitant medications
- 2.1.3 Efficacy endpoints
- 2.1.3.1 Primary efficacy endpoint(s)
- 2.1.3.2 Secondary efficacy endpoint(s)
- 2.1.3.3 Other efficacy endpoint(s)
- 2.1.4 Safety endpoints
- 2.1.4.1 Hypoglycemia
- 2.1.4.2 Adverse events variables
- 2.1.4.3 Deaths
- 2.1.4.4 Laboratory safety variables
- 2.1.4.5 Vital signs variables
- 2.1.4.6 Physical examination

INTERIM ANALYSIS

| 2.1.4.7 | Electrocardiogram variables |
|---|---|
| 2.1.5 | Pharmacokinetic variables |
| 2.2 | DISPOSITION OF PATIENTS |
| 2.2.1 | Randomization and drug dispensing irregularities |
| 2.3 | ANALYSIS POPULATIONS |
| 2.3.1 | Efficacy populations |
| 2.3.1.1 | Intent-to-treat population |
| 2.3.2 | Safety population |
| 2.3.3 | Pharmacokinetic population |
| 2.4 | STATISTICAL METHODS |
| 2.4.1 | Demographics and baseline characteristics |
| 2.4.2 | Prior or concomitant medications |
| 2.4.3 | Extent of investigational medicinal product exposure and compliance |
| 2.4.3.1 | Extent of investigational medicinal product exposure |
| 2.4.3.2 | Compliance |
| 2.4.4 | Analyses of efficacy endpoints |
| 2.4.4.1 | Analysis of primary efficacy endpoint |
| 2.4.4.2 | Analyses of secondary efficacy endpoints |
| 2.4.4.3 | Analyses of other efficacy endpoints |
| 2.4.4.4 | Multiplicity issues |
| 2.4.5 | Analyses of safety data |
| 2.4.5.1 | Analyses of hypoglycemia |
| 2.4.5.2 | Analyses of adverse events |
| 2.4.5.3 | <u>Deaths</u> |
| 2.4.5.4 | Analyses of laboratory variables |
| 2.4.5.5 | Analyses of vital sign variables |
| 2.4.5.6 | Analyses of electrocardiogram variables |
| 2.4.5.7 | Analyses of physical examination variables |
| 2.4.6 | Analyses of pharmacokinetic variables |
| 2.5 | DATA HANDLING CONVENTIONS |
| 2.5.1 | General conventions |
| 2.5.2 | Data handling conventions for secondary efficacy variables |
| 2.5.3 | Missing data |
| 2.5.4 | Windows for time points /Measurements for analyses |
| 2.5.5 | Unscheduled visits |
| 2.5.6 | Pooling of centers for statistical analyses |
| 2.5.7 | Statistical technical issues |

- 4 DATABASE LOCK
- 5 SOFTWARE DOCUMENTATION
- 6 REFERENCES
- 7 LIST OF APPENDICES
- APPENDIX A POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES CRITERIA
- APPENDIX B LIST OF PTS FOR SELECT EOSIS (MEDDRA V22.0)
- APPENDIX C SUMMARY OF STATISTICAL ANALYSES
- APPENDIX D STUDY FLOW CHART

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

AEs: adverse events

AESI: adverse events of special interest

ALT: alanine aminotransferase
ANCOVA: analysis of covariance
AST: aspartate aminotransferase
BLOQ: below limit of quantification
ATC: anatomical therapeutic chemical

BMI: body mass index BUN: blood urea nitrogen

CEC: clinical endpoint committee

CI: confidence interval

CMH: Cochran-Mantel-Haenszel CV: cardiovascular, cardiovascular

DBP: diastolic blood pressure

DCCT: diabetes control and complications trial

DILI: drug-induced liver injury
DMC: Data Monitoring Committee

ECG: electrocardiogram

e-CRF: electronic case report form

eGFR: estimated glomerular filtration rate

EMA/PRAC: European Medicines Agency/ Pharmacovigilance Risk Assessment Committee

EOSI: events of special interest

EOT: end of treatment

FPG: fasting plasma glucose

Gd: glibenclamide GdMR: glibenclamide MR

Gp: glipizide
GpXL: glipizide XL
Gz: gliclazide
GzMR: gliclazide MR
HbA1c: hemoglobin A1c
HLGT: high level group term
HLT: high level term

heart rate

IFCC: International Federation of Clinical Chemistry and Laboratory Medicine

IMP: investigational medicinal product INN: international nonproprietary name IRT: interactive response technology

ITT: intent-to-treat
KM: Kaplan-Meier
LLT: lower level term

HR:

MACE: major adverse cardiovascular events

Date of Issue: 19 February 2020 Covance Study ID:000000154257 Lexicon Pharmaceuticals Protocol No. EFC14835

MAR: missing at random

modification of diet in renal disease MDRD:

MedDRA: Medical Dictionary for Regulatory Activities

multiple imputation MI: missing not at random MNAR:

noninvestigational medicinal product NIMP:

PCSA: potentially clinically significant abnormality

PD: pharmacodynamic pharmacokinetic PK: PT: preferred term

SAE: serious adverse events SBP: systolic blood pressure standard deviation SD: system organ class SOC: T2D: type 2 diabetes mellitus

TEAE: treatment-emergent adverse event

upper limit of normal ULN:

WHO-DD: World Health Organization-Drug Dictionary

## 1 OVERVIEW AND INVESTIGATIONAL PLAN

#### 1.1 STUDY DESIGN AND RANDOMIZATION

This is a Phase 3, multicenter and multinational, randomized, double-blind, placebo-controlled, parallel-group study. Patients will be randomly assigned 1:1 to the following 2 treatment groups

- Sotagliflozin 400 mg.
- Placebo.

All patients will have a Screening Period comprised of an up to 2-week Screening Phase and a 2-week, single-blind placebo Run-in Phase prior to randomization. Following randomization, patients will have a 26-week, double-blind Core Treatment Period, a 53-week double-blind Extension Period, and a 2-week post-treatment Follow-up period to collect safety information (patients who prematurely discontinue the study treatment are expected to continue in the study).

At the end of the screening period, eligible patients will be centrally randomized (using permuted block randomization schedule) via an Interactive Response Technology (IRT). The randomization will be stratified by

- Hemoglobin A1c (HbA1c) at Screening ( $\leq 8.5\%$ , > 8.5%).
- Metformin use at Screening (Yes, No).
- Systolic blood pressure (SBP) at Screening (<130 mmHg, ≥130 mmHg).</li>

It is anticipated to randomize a total of approximately 500 patients.

#### 1.2 OBJECTIVES

#### 1.2.1 Primary objectives

The primary objective of this study is to demonstrate the superiority of sotagliflozin 400 mg versus placebo on HbA1c reduction at Week 26 in patients with type 2 diabetes mellitus (T2D) who have inadequate glycemic control with a sulfonylurea alone or in combination with metformin.

## 1.2.2 Secondary objectives

- To compare sotagliflozin 400 mg versus placebo for:
  - Change from Baseline in fasting plasma glucose (FPG) at Week 26,
  - Change from Baseline in body weight at Week 26,
  - Change from Baseline in SBP at Week 12 for patients with baseline SBP ≥130 mmHg,

- Change from Baseline in SBP at Week 12 for all patients,
- Proportion of patients with HbA1c <6.5%, <7.0% at Week 26.
- To evaluate the safety of sotagliflozin 400 mg versus placebo throughout the 79-week trial.

#### 1.2.3 Other objectives

- To compare sotagliflozin versus placebo based on other blood pressure endpoints.
- To compare sotagliflozin versus placebo with respect to change from Baseline on the following endpoints:
  - Estimated glomerular filtration rate (eGFR),
  - Reduction in body weight by  $\geq 2\%$ ,  $\geq 5\%$ , and  $\geq 10\%$ .
- To compare sotagliflozin versus placebo for:
  - Change from Baseline in HbA1c at Week 79,
  - Change from Baseline in FPG at Week 79,
  - Change from Baseline in body weight at Week 79.
- To compare the use of rescue medications for hyperglycemia in the sotagliflozin and placebo treatment groups.
- To assess plasma concentrations of sotagliflozin and its 3-O-glucuronide metabolite.

### 1.3 DETERMINATION OF SAMPLE SIZE

The sample size/power calculations are based on the primary variable, change from Baseline to Week 26 in HbA1c. Assuming a common standard deviation (SD) of 1.2% and using a 2-sided test at a 0.05  $\alpha$ -level, 250 patients per arm will have 99% power to detect a treatment difference of 0.6% in mean HbA1c change from Baseline to Week 26 between sotagliflozin 400 mg and placebo.

The number of patients taking a sulfonylurea and metformin will be limited to 330 patients, to ensure sufficient numbers of sulfonylurea monotherapy patients.

## 1.4 STUDY PLAN



The study flowchart can be found in Appendix D.

### 1.5 MODIFICATIONS TO THE STATISTICAL SECTION OF THE PROTOCOL

This section summarizes major changes to the protocol statistical section with emphasis on changes after study start (after the first patient was enrolled).

The protocol history table below gives the timing, rationale, and key details of major changes to the protocol statistical section.

The first patient was enrolled on Feb 24, 2017. There were no planned interim analyses.

Table 1 - Protocol amendment statistical changes

| Amendment<br>Number | Date<br>Approved | Rationale | Description of statistical changes |
|---|---|---|---|
| 2 | 20-Dec-2017 | 5 half-lives of sotagliflozin prolonged<br>to 10 days considering patients with<br>moderate renal dysfunction | 5 half-lives of IMP updated from 5 days to 10 days; TEAE period updated accordingly |
| 2 | 20-Dec-2017 | Baseline eGFR defined as<br>recommended by CDISC Therapeutic<br>Area Data Standards User Guide for<br>Diabetic Kidney Disease | For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP. |
| 2 | 20-Dec-2017 | The effect in body weight is<br>considered more closely associated<br>with the planned indication | Change in the order of secondary objectives, endpoints and multiplicity considerations |
| 2 | 20-Dec-2017 | Urgent coronary revascularization not<br>adjudicated by CEC to be consistent<br>with outcome trials | Urgent coronary revascularization not included in adjudication related analyses |
| 2 | 20-Dec-2017 | AE leading to study discontinuation is<br>less clinically relevant than AE<br>leading to treatment discontinuation | Delete AEs leading to discontinuation from the study from safety endpoints |
| 2 | 20-Dec-2017 | To understand treatment effects over the entire study duration | Several objectives/endpoints "blood pressure<br>endpoints at Week 26 and Week 79, HbA1c,<br>FPG and body weight endpoints at Week 79"<br>were added |

## 1.6 STATISTICAL MODIFICATIONS MADE IN THE STATISTICAL ANALYSIS PLAN

The statistical analysis plan history table below gives the timing, rationale, and key details for major changes to the statistical analysis features in the statistical analysis plan. Changes also incorporated in a protocol amendment are cross-referenced to Table 1.

Date of Issue: 19 February 2020 Covance Study ID:000000154257

Table 2 - Statistical analysis plan statistical changes

| SAP | | | |
|---|---|---|---|
| version<br>number | Date<br>approved | Rationale | Description of statistical changes |
| 1 | 07-Aug-2018 | 5 half-lives of sotagliflozin prolonged to<br>10 days considering patients with<br>moderate renal dysfunction | 5 half-lives of IMP updated from 5 days to 10 days; TEAE period updated accordingly* |
| 1 | 07-Aug-2018 | Baseline eGFR defined as<br>recommended by CDISC Therapeutic<br>Area Data Standards User Guide for<br>Diabetic Kidney Disease | For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP* |
| 1 | 07-Aug-2018 | The effect in body weight is considered<br>more closely associated with the<br>planned indication | Change in the order of secondary objectives, endpoints and multiplicity considerations* |
| 1 | 07-Aug-2018 | Urgent coronary revascularization not<br>adjudicated by CEC to be consistent<br>with outcome trials | Urgent coronary revascularization not included in adjudication related analyses* |
| 1 | 07-Aug-2018 | AE leading to study discontinuation is<br>less clinically relevant than AE leading<br>to treatment discontinuation | Delete AEs leading to discontinuation from the study from safety endpoints* |
| 1 | 07-Aug-2018 | To understand treatment effects over the entire study duration | Several objectives/endpoints "blood pressure<br>endpoints at Week 26 and Week 79, HbA1c,<br>FPG and body weight endpoints at Week 79"<br>were added* |
| 1 | 07-Aug-2018 | Clarification on EOSI renal events | Details specified on renal events to be consistent with outcome studies in Section 2.1.4.2. |
| 1 | 07-Aug-2018 | | |
| 1 | 07-Aug-2018 | | |
| 1 | 07-Aug-2018 | Updating the wording to be consistency with CEC charter | Unstable angina leading to hospitalization<br>changed to Unstable angina requiring<br>hospitalization |
| 2 | 03-Jun-2019 | | |
| 2 | 03-Jun-2019 | Number of iterations for multiple imputation was changed | Number of iterations for multiple imputation was changed from 10 000 to 2000 |
| 2 | 03-Jun-2019 | Wording change to be consistent with<br>CEC charter | "Heart failure leading to hospitalization" changed to "Heart failure requiring hospitalization" |
| 2 | 03-Jun-2019 | MedDRA version and dictionary<br>updated | MedDRA version was updated to V22.0 and list<br>of PTs for selected EOSI were updated |
| 3 | This version | | |

| SAP<br>version<br>number | Date<br>approved | Rationale | Description of statistical changes |
|---|---|---|---|
| 3 | This version | | |
| 3 | This version | | |
| 3 | This version | | |
| 3 | This version | | |

<sup>\*</sup> Change made in Protocol Amendment 2 dated 20-Dec-2017.

## 2 STATISTICAL AND ANALYTICAL PROCEDURES

#### 2.1 ANALYSIS ENDPOINTS

## 2.1.1 Demographic and baseline characteristics

The baseline value for all variables (with the exception of serum creatinine and eGFR) is defined as the last available value before the first dose of double-blind investigational medicinal product (IMP), or the last available value prior to randomization for patients who were randomized but never exposed to IMP.

For serum creatinine and eGFR, the baseline value is defined as the average of all values before the first dose of double-blind IMP for those randomized and exposed or before randomization for those who were randomized but never exposed to IMP.

Baseline safety and efficacy parameters are presented along with the summary statistics for safety and efficacy sections (Section 2.4.4 and Section 2.4.5).

## Demographic characteristics

Demographic characteristics to be summarized are:

- Age (years) derived as: (Year of informed consent Year of birth).
- Age categories:  $(<50, \ge 50 \text{ to } < 65, \ge 65 \text{ to } < 75, \ge 75 \text{ years})$ .
- Gender (Male, Female).
- Race (White, Black or African American, Asian, American Indian or Alaska native, Native Hawaiian or other pacific islander, Multiple, Unknown).
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Unknown).
- HbA1c (%) at screening visit.
- Randomization strata of HbA1c (\le 8.5\%, \rightarrow 8.5\%) at screening (data from IRT).
- Randomization strata of metformin use (Yes, No) at screening (data from IRT).
- Mean SBP at screening.
- Randomization strata of SBP (<130 mmHg, ≥130 mmHg) at screening (data from IRT).</li>
- Baseline body mass index (BMI) (kg/m<sup>2</sup>) derived as: (Weight in kg)/(Height in meters)<sup>2</sup>.
- Baseline BMI categories (<30, ≥30 kg/m²).</li>
- Country.

### Disease characteristics at screening or baseline

## Disease history includes:

- Duration of diabetes (years) derived as: (Date of informed consent Date of diagnosis of diabetes + 1)/365.25.
- Duration of diabetes categories:  $(<10, \ge 10 \text{ years})$ .
- Age at diagnosis of diabetes (years): (Year of diagnosis of diabetes Year of birth).
- Metformin use at screening (Yes, No).
- Duration of metformin treatment (for those patients who used metformin at screening) (years): (date of informed consent date of first intake of metformin +1)/365.25.
- Daily dose of metformin (mg) at baseline (for those patients who used metformin at screening).
- Categorized daily dose of metformin at baseline for those patients who used metformin at screening (<1500, ≥1500 to <2500, ≥2500 mg).
- Duration of sulfonylurea treatment (years): (date of informed consent date of first intake of sulfonylurea +1)/365.25.
- Sulfonylurea at screening by international nonproprietary name (INN) and formulation.
- Daily dose of sulfonylurea at baseline by INN and formulation.
- Categorized daily dose of sulfonylurea at baseline by INN:
  - Glibenclamide (Gd) and Glibenclamide MR (GdMR):
    - <10 mg/day (Gd) or <6 mg/day (GdMR),
    - $\geq 10 \leq 20 \text{ mg/day (Gd) or } \geq 6 \leq 12 \text{ mg/day (GdMR)},$
    - $\geq$ 20 mg/day (Gd) or  $\geq$ 12 mg/day (GdMR).
  - Gliclazide (Gz) and Gliclazide MR (GzMR):
    - <160 mg/day (Gz) or <60 mg/day (GzMR),
    - $\ge 160 \le 320 \text{ mg/day (Gz) or } \ge 60 \le 120 \text{ mg/day (GzMR)},$
    - >320 mg/day (Gz) or >120 mg/day (GzMR).
  - Glimepiride:
    - <4 mg/day,</li>
    - ≥4 ≤8 mg/day,
    - >8 mg/day.
  - Glipizide (Gp) and Glipizide XL (GpXL):
    - <20 mg/day (Gp) or <10 mg/day (GpXL),</li>
    - $\geq$ 20  $\leq$ 40 mg/day (Gp) or  $\geq$ 10  $\leq$ 20 mg/day (GpXL),

- Date of Issue: 19 February 2020 Covance Study ID:000000154257
- >40 mg/day (Gp) or >20 mg/day (GpXL).
- Gliquidone:
  - <90 mg/day,</p>
  - $\ge 90 \le 180 \text{ mg/day},$
  - >180 mg/day.
- Baseline diabetic microvascular complications (Yes, No) (ie, diabetic retinopathy, diabetic neuropathy, diabetic nephropathy, diabetic peripheral neuropathy (sensory or motor), diabetic autonomic neuropathy, and diabetic foot infection).
- eGFR at screening (mL/min/1.73m<sup>2</sup>).
- eGFR categories at screening (<15 mL/min/1.73m<sup>2</sup> [End stage renal disease], ≥15 to <30 mL/min/1.73m<sup>2</sup> [Severe decrease in GFR], ≥30 to <60 mL/min/1.73m<sup>2</sup> [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m<sup>2</sup> [Mild decrease in GFR], and ≥90 mL/min/1.73m<sup>2</sup> [Normal]).
- Prior antihypertensive medication identified by therapeutic class as agents acting on the renin-angiotensin system, beta blocking agents, diuretics (a sub-category: loop diuretics identified by pharmacological class as high-ceiling diuretics), calcium channel blockers, and antihypertensives according to World Health Organization-Drug Dictionary (WHO-DD).

## Medical or surgical history

Medical history and medical findings include:

- Physical examination.
- Medical or surgical history.
- Medical history cardiovascular.
- Surgical history amputation.
- Alcohol habits.
- Tobacco smoking habits.

Medical and surgical history will be coded to a "lower level term (LLT)", "preferred term (PT)", "high level term (HLT)", "high level group term (HLGT)", and associated primary "system organ class (SOC)" using the version of Medical Dictionary for Regulatory Activities (MedDRA) currently in effect at Covance at the time of database lock.

Any technical details related to computation, dates, and imputations for missing dates are described in Section 2.5.

#### 2.1.2 Prior or concomitant medications

All medications taken within 3 months before the screening visit (any time for prior SGLT2) and until the end of the study are to be reported in the electronic case report form (e-CRF).

All medications will be coded using the World Health Organization-Drug Dictionary WHO-DD using the version currently in effect at Covance at the time of database lock.

- Prior medications are those the patient used prior to first administration of the doubleblind IMP. Prior medications can be discontinued before first administration or can be ongoing during treatment phase.
- Concomitant medications are any treatments received by the patient concomitantly to the IMP, from the 1<sup>st</sup> administration of double-blind IMP to the date of last administration + 10 days. A given medication can be classified both as a prior medication and as a concomitant medication.
- Posttreatment medications are those the patient took in the period running from the 11th day after the last administration of double-blind IMP up to the end of the study.

Background sulfonylurea and metformin are considered as noninvestigational medicinal products (NIMP). Sulfonylurea and metformin (commercial formulations) will be administered orally according to the locally approved label.

Any technical details related to computation, dates, imputation for missing dates are described in Section 2.5.

#### 2.1.2.1 Rescue therapy

Except for SGLT2 inhibitors and additional metformin and sulfonylurea, any approved medication(s) including oral antidiabetic drugs, GLP-1 receptor agonists, or insulin can be prescribed at the Investigator's discretion to treat the hyperglycemia. Metformin will also be permitted for patients on sulfonylurea only at Screening. Rescue therapy is considered a NIMP.

## 2.1.2.2 Prohibited prior and concomitant medications

During the study treatment period, the following medications are prohibited:

- Initiation of any antidiabetic agents, including oral or injectable antihyperglycemic agents other than the IMP before the rescue therapy.
  - Note: short term use (<10 consecutive days) of the prohibited medication, eg, short-acting insulin for treatment of acute illness or surgery is allowed.
- Systemic use of glucocorticoids for more than 10 consecutive days (topical, ophthalmic, nasal spray or inhaled applications are allowed).
- Initiation of any weight loss drugs (eg, phentermine, orlistat).

Investigational medicinal products in any other clinical study.

SGLT2 inhibitors (eg, canagliflozin, dapagliflozin, or empagliflozin), additional sulfonylurea and metformin are not allowed for rescue or post IMP therapy until the end of study.

Reduction of digoxin dose should be considered because sotagliflozin acts as a weak P-glycoprotein inhibitor and increases systemic exposure to digoxin.

Other medications which are unlikely to interfere with the pharmacokinetic (PK) or pharmacodynamic (PD) of the IMP or confound interpretation of the study endpoints are allowed as needed following discussion between the Investigator and the Sponsor. However, doses of chronically administered medicines should be kept fixed during the trial if at all possible.

After premature permanent discontinuation of the IMPs, any treatments (other than SGLT2 inhibitors) are permitted, as deemed necessary by the Investigator.

The dose of all antihypertensive agents should be kept constant during the 12 weeks following randomization and no antihypertensive agents should be added or withdrawn for the 12 weeks following randomization unless it is considered necessary for safety reasons.

## 2.1.3 Efficacy endpoints

All efficacy measurements collected during the study will be considered for analyses, including those obtained after IMP discontinuation or introduction of rescue therapy (see Section 2.5.4).

HbA1c, FPG, serum creatinine, eGFR are measured/calculated in a central laboratory (see study flowchart in D). Body weight, SBP and diastolic blood pressure (DBP) (see Section 2.1.4.5) are measured at on-site visits by the investigator. Patients requiring rescue are identified as those with the reason for treatment ticked "rescue therapy" in e-CRF "Medication" page.

Efficacy variables will be summarized in both standard international units and conventional units when applicable.

#### 2.1.3.1 Primary efficacy endpoint(s)

• Change from Baseline to Week 26 in HbA1c (%).

#### 2.1.3.2 Secondary efficacy endpoint(s)

- Change from Baseline to Week 26 in FPG.
- Change from Baseline to Week 26 in body weight.
- Change from Baseline to Week 12 in SBP for patients with baseline SBP ≥130 mmHg.
- Change from Baseline to Week 12 in SBP for all patients.
- Proportion of patients with HbA1c <6.5%, <7.0% at Week 26.</li>

## 2.1.3.3 Other efficacy endpoint(s)

- Change from Baseline to Week 12 in SBP for patients with baseline SBP <130 mmHg.</li>
- Proportion of patients with reduction in body weight by ≥2%, ≥5%, and ≥10% from Baseline.
- Change from Baseline to Week 12 in DBP.
- Proportion of patients achieving SBP <130 mmHg for those with baseline SBP ≥130 mmHg.</li>
- Proportion of patients achieving DBP <80 mmHg for those with baseline DBP ≥80 mmHg.</li>
- Proportion of patients requiring rescue for hyperglycemia.
- Change from Baseline in:
  - Serum creatinine,
  - eGFR.
- Change from Baseline to Week 79 in HbA1c.
- Change from Baseline to Week 79 in FP.
- Change from Baseline to Week 26 in SBP for all patients and for patients with baseline SBP ≥130 mmHg.
- Change from Baseline to Week 79 in SBP for all patients and for patients with baseline SBP ≥130 mmHg.
- Change from Baseline to Week 79 in body weight.

## 2.1.4 Safety endpoints

The safety analysis will be based on the reported adverse events (AEs), hypoglycemia, and other safety information, such as clinical laboratory data, vital signs, electrocardiogram (ECG), and physical examination, etc.

## Observation period

The observation period will be divided into 4 epochs:

- The **screening** epoch is defined as the time from the signed informed consent date up to the first administration of the double-blind IMP.
- The **treatment** epoch is defined as the time from the first administration of the double-blind IMP to the last administration of the double-blind IMP. This epoch includes the 26-week double-blind core treatment period and the 53-week double-blind extension treatment period. The core treatment period is the time from the first administration of double-blind IMP to the last administration of double-blind IMP on or before Visit 9/Week 26 (or Day 182 if Visit 9/Week 26 date is missing).

 The residual treatment epoch is defined as the time from the last administration of the double-blind IMP up to 10 days (1 day for hypoglycemia) after the last administration of double-blind IMP.

The treatment-emergent adverse event (TEAE) period will include both treatment and residual treatment epochs (See the TEAE period for the core treatment period in Section 2.5.4).

• The **posttreatment** epoch is defined as the period of time starting the day after the end of the TEAE period up to the last protocol-planned visit or the resolution/stabilization of all serious adverse events (SAE), adverse events of special interest (AESI) and events of special interest (EOSI), whichever is later.

The on-study observation period is defined as the time from start of double-blind treatment until the end of the study (defined as the last scheduled visit for those who completed the study and the date collected on e-CRF page "Completion of End of Study/Follow-up" for those who did not complete the study).

The post-study observation period is defined as the time from the day after the end of the study until the resolution/stabilization of all SAE, AESI and EOSI if applicable.

## 2.1.4.1 Hypoglycemia

Hypoglycemia will be identified as events recorded on the dedicated e-CRF "Hypoglycemic event information" page, and will be categorized as follows (see study protocol for further details):

#### Severe hypoglycemia

Severe hypoglycemia is an event requiring assistance of another person to actively administer carbohydrate, glucagon, intravenous glucose or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure, unconsciousness or coma.

Self-monitored plasma glucose values may not be available, but neurological recovery attributable to the restoration of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.

Severe hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- To the question "Countermeasure Administration", ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and
- 2. To the question "Were Symptoms Present", ticked "Yes".

#### Documented symptomatic hypoglycemia

Documented symptomatic hypoglycemia is an event during which typical symptoms of hypoglycemia accompanied by a measured plasma glucose concentration of  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL).

Clinical symptoms that are considered to result from a hypoglycemic episode are eg, increased sweating, nervousness, asthenia/weakness, tremor, dizziness, increased appetite, palpitations, headache, sleep disorder, confusion, seizures, unconsciousness, or coma.

Documented symptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as:

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and,
- 2. To the question "Were Symptoms Present", ticked "Yes", and,
- 3. With a plasma glucose value before countermeasure  $\leq$  3.9 mmol/L ( $\leq$  70 mg/dL).

## Asymptomatic hypoglycemia

Asymptomatic hypoglycemia is an event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration  $\leq$  3.9 mmol/L ( $\leq$ 70 mg/dL).

Asymptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as:

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and,
- 2. To the question "Were Symptoms Present", ticked "No", and,
- 3. With a plasma glucose value before countermeasure  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL).

## Probable symptomatic hypoglycemia

Probable symptomatic hypoglycemia is an event during which symptoms of hypoglycemia are not accompanied by a plasma glucose determination, (but that was presumably caused by a plasma glucose concentration  $\leq$ 3.9 mmol/L [ $\leq$ 70 mg/dL]), ie, symptoms treated with oral carbohydrate without a test of plasma glucose.

Probable symptomatic hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance", and,
- 2. To the question "Were Symptoms Present", ticked "Yes", and,
- 3. With no plasma glucose value before countermeasure, and,
- 4. To the question "Did this countermeasure lead a significant improvement or prompt recovery?", ticked "Yes".

### Relative hypoglycemia

Relative hypoglycemia, recently termed "pseudo hypoglycemia", is an event during which the patient reports typical symptoms of hypoglycemia, and interprets the symptoms as indicative of hypoglycemia, but with a measured plasma glucose concentration >3.9 mmol/L (>70 mg/dL).

Relative hypoglycemia is identified in e-CRF "Hypoglycemic event information" page as those documented as,

- 1. To the question "Countermeasure Administration", NOT ticked the option "Subject was Not Capable of Treating Self and Required Assistance",
- 2. To the question "Were Symptoms Present", ticked "Yes", and,
- 3. With a plasma glucose value before countermeasure >3.9 mmol/L (>70 mg/dL).

In addition of the threshold of  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL), hypoglycemia episodes with a plasma glucose of  $\leq$ 3.0 mmol/L ( $\leq$ 54 mg/dL) will be analyzed separately.

Any hypoglycemic event fulfilling the criteria of a SAE or leading to unconsciousness, coma, or seizure will also be recorded as a SAE (Section 2.1.4.2).

#### 2.1.4.2 Adverse events variables

#### AE observation period

- **Pretreatment AEs** are AEs that developed or worsened or became serious from the signed informed consent date up to first administration of double-blind IMP.
- TEAEs are AEs that developed or worsened or became serious during the TEAE period.
- Posttreatment AEs are AEs that developed or worsened or became serious during the
  posttreatment period.

All AEs (including SAEs, AESI and EOSI) will be coded to a LLT, PT, HLT, HLGT, and associated SOC using the version of MedDRA currently in effect at Covance at the time of database lock.

The occurrence of AEs (including SAEs, AESI and EOSI) will be recorded from the time of signed informed consent until the end of the study (see Section 2.1.4) or the resolution/stabilization of all SAE, AESI and EOSI.

#### **AESI** include

- Pregnancy.
- Symptomatic overdose with IMP/NIMP.
- Alanine aminotransferase (ALT) increase > 3 × upper limit of normal (ULN).

#### **EOSI** include

- Major adverse cardiovascular events (MACE [cardiovascular death, myocardial infarction, or stroke]) and other specific cardiovascular (CV) events (eg, heart failure requiring hospitalization).
- Severe hypoglycemia.
- Genital mycotic infections (to include vulvovaginal candidiasis in females and candida balanitis in males).
- Urinary tract infection.
- Clinically relevant volume depletion and events related/possibly related to volume depletion.
- Diarrhea.
- Pancreatitis.
- Bone fractures.
- Venous thrombotic events, to include deep venous thrombosis and thromboembolism (to include pulmonary embolism).
- Diabetic ketoacidosis.
- Renal events, to include 50% decline in eGFR, end stage kidney disease, renal death.
- Malignancies of special interest (breast, bladder, renal cell, Leydig cell, pancreatic, prostate, and thyroid cancer).
- AE leading to an amputation.

A Clinical Endpoint Committee (CEC) will, in a blinded manner, review and adjudicate all deaths, myocardial infarction, stroke, unstable angina requiring hospitalization, and heart failure requiring hospitalization, selected renal events, bone fracture, and diabetic ketoacidosis.

Two independent committees will review safety events that require ongoing monitoring to ensure timing protocol amendments in case a safety signal is identified. These events are: 1) potential cases of drug-induced liver injury (DILI), and 2) cases of amputations. The two committees will review the cases in a treatment-blinded manner and will present their assessment to the DMC.

AESI and EOSI will be identified based on criteria in Table 3.

Table 3 - Criteria for AESI and EOSI

| | Table 3 - Criteria for AESI and EOSI |
|---|---|
| AE Grouping | Criteria |
| AESI | |
| Pregnancy | e-CRF "Pregnancy" |
| Symptomatic overdose with IMP/NIMP | "Overdose of IMP" or "Overdose of NIMP" checked and "Symptomatic overdose" checked in e-CRF "Overdose" |
| ALT increase >3 × ULN | e-CRF "ALT increase" |
| EOSI adjudicated | |
| Cardiovascular death | Positively adjudicated by CEC: "Cardiovascular" or "Undetermined" as the primary cause of death |
| Myocardial infarction, Unstable<br>Angina requiring hospitalization | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of an MI for this study?", or Yes to the question "If event is not an MI, does the event meet the definition of an UA Requiring admission to hospital or emergency room, for this study?" |
| Stroke | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of a Stroke for this study?" |
| Heart failure requiring hospitalization | Positively adjudicated by CEC: Yes to the question "Does the event meet the definition of a Heart Failure Event for this study?" |
| Bone fractures | Positively adjudicated by CEC: Yes to the question "Did the Fracture occur?" |
| Diabetic ketoacidosis | Positively adjudicated by CEC: Yes to the question "Does this event meet the criteria to be a DKA event?" |
| EOSI Renal events where select ev | vents adjudicated |
| Sustained ≥50% decrease in eGFR | (1) For ≥50% decrease in eGFR from baseline, |
| | (1a) confirmed ≥50% decrease in GFR for ≥30 days with no reversible cause as recorded in e-CRF "eGFR decrease", OR |
| | (1b) positively adjudicated by CEC: Yes to the question "Does the subject meet the criteria of CKD progression" for ≥50% decrease in eGFR. |
| Sustained eGFR <15 mL/min/1.73 | (2) For eGFR <15 mL/min/1.73 m2, |
| m2 | (2a) confirmed eGFR <15 mL/min/1.73 m2 for $\geq$ 30 days with no reversible cause as recorded in e-CRF "eGFR decrease", OR |
| | (2b) positively adjudicated by CEC: Yes to the question "Does the subject meet the criteria of CKD progression". |
| Chronic dialysis | (3) For dialysis, (3a) dialysis lasted for ≥90 days (eg, end date – start date+ 1 ≥90) as recorded in e-CRF "Renal Event – Dialysis", OR (3b) positively adjudicated by CEC: Yes to the question ". Does the subject meet the criterio for ESRD" |
| Renal transplant* | criteria for ESRD". (4) "Renal transplant" captured in e-CRF "Other procedure form", where adjudication is not required. PTs of Renal transplant (10038533), Renal and pancreas transplant (10052278), Renal and liver transplant (10052279) based on MedDRA v22.0. |
| Renal death | (5) Renal death as positively adjudicated by CEC: "Death - Non-Cardiovascular (Renal)" as the primary cause of death |

| AE Grouping | Criteria |
|---|---|
| EOSI not adjudicated* | |
| Severe hypoglycemia | Algorithm specified in Section 2.1.4.1 based on e-CRF "Hypoglycemic Events" |
| Genital mycotic infections | PTs in Appendix B |
| Urinary tract infections | PTs in Appendix B |
| Clinically relevant volume depletion and events related/possibly related to volume depletion | PTs in Appendix B |
| Diarrhea | Narrow search on "Noninfectious diarrhoea (SMQ)" [20000218] plus the following PTs (MedDRA v22.0): Gastroenteritis (10017888), Antidiarrhoeal supportive care (10055660), Enteritis (10014866), Enteritis leukopenic (10014877), Enterocolitis (10014893), Enterocolitis haemorrhagic (10014896) |
| Pancreatitis | PTs in Appendix B |
| Venous thrombotic events | PTs in Appendix B |
| Malignancies of special interest | Breast cancer: Narrow search on "Breast cancer: Narrow search on "Breast neoplasms, malignant and unspecified (SMQ)" [20000149] |
| | Prostate cancer: Narrow search on "Prostate neoplasms, malignant and unspecified (SMQ)" [20000152] |
| | Leydig-cell cancer: PTs of Leydig cell tumour of the testis (10024407) and Ovarian Sertoli-<br>Leydig cell tumour (10073270) based on MedDRA v22.0 |
| | Thyroid cancer: PTs in Appendix B |
| | Renal cell cancer: PTs in Appendix B |
| | Pancreatic cancer: PTs in Appendix B |
| | Bladder cancer: PTs in Appendix B |
| EOSI AE leading to an amputation | 1 |
| AE leading to an amputation | "AE Correction" as the reason for amputation in e-CRF "Other Procedures related to Amputation" |
| AE potentially leading to an amputation * | PTs in Appendix B |

<sup>\*</sup> Search terms will be updated using the MedDRA version currently in effect at Covance at the time of database lock for EOSI identified by them.

#### 2.1.4.3 Deaths

The deaths observation period are per the observation periods defined above.

- Death on-study: deaths occurring during the on-study observation period.
- Death on-treatment: deaths occurring during the TEAE period.
- Death post-study: deaths occurring after the end of the study.

<sup>\*</sup> AE potentially leading to an amputation: not belong to the EOSI list defined in protocol, the item is included and analyzed due to their relevance in regards to lower limb complications and amputations as a requirement from health authorities..

## 2.1.4.4 Laboratory safety variables

Clinical laboratory data consists of blood analysis (including hematology, clinical chemistry, amylase, lipase and lipid profile) and urinalysis. Clinical laboratory values will be summarized in both standard international units and conventional units when applicable.

Blood samples for clinical laboratories will be collected at designated visits (see study flowchart in D). The following laboratory data will be measured at a central laboratory:

- Hematology
  - Red blood cells and platelets: hemoglobin, hematocrit, red blood cell, platelets count,
  - White blood cells: white blood cell, neutrophils, lymphocytes, monocytes, basophils, eosinophils.
- Clinical chemistry
  - Metabolism: glucose (serum), creatine phosphokinase (CPK),
  - Electrolytes and minerals: sodium, potassium, chloride, bicarbonate (ie, carbon dioxide), calcium, phosphorus, magnesium,
  - Renal function: blood urea nitrogen (BUN), creatinine, uric acid,
  - Liver function: total protein, albumin, ALT, aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin, Lactic acid dehydrogenase (LDH).
- Lipid parameters (fasting): total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C) (calculated by Friedwald equation, See Section 2.5.1), Non-HDL-C (calculated as the difference between TC and HDL-C), triglycerides (TG).
- Pancreatic enzymes: lipase, amylase.

Urine samples will be collected at designated visits (see study flowchart in . The following laboratory data will be measured at a central laboratory:

- Urine dipstick includes: specific gravity, pH, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase.
- Urine microscopy includes, but is not limited to: detection of formed cellular elements, casts, bacteria, yeast, parasites, and crystals in centrifuged urine sediment.

Serum glucose will be presented as efficacy parameters in Section 2.4.4. For creatinine and calculated eGFR, Potentially Clinically Significant Abnormality (PCSA) summaries will be presented in the safety section while descriptive summaries in the efficacy section.

Technical formulas are described in Section 2.5.1.

## 2.1.4.5 Vital signs variables

Vital signs include: heart rate (HR), systolic and diastolic blood pressure, temperature, and respiratory rate. They will be performed after the patient has been seated for at least 5 minutes. Blood pressure and HR will be assessed 3 times with at least 1 minute between each measurement. The mean of the 3 measurements will be analyzed for each vital sign variable (HR, SBP, and DBP).

### 2.1.4.6 Physical examination

A complete physical exam will be performed at Visit 1 (Screening), Visit 9 (Week 26) and Visit 13 (Week 79). "Normal", "Abnormal" or "Not done" as determined by the Investigator will be reported in the e-CRF by body system.

## 2.1.4.7 Electrocardiogram variables

12-lead ECGs will be performed at Visit 1 (Screening), Visit 9 (Week 26), and Visit 13(Week 79). ECG status of "normal" or "abnormal" will be reported in the e-CRF as determined by the investigator.

#### 2.1.5 Pharmacokinetic variables

Pharmacokinetic variables include the plasma concentration of sotagliflozin and its 3-O-glucuronide metabolite in the sotagliflozin 400 mg group.

#### 2.2 DISPOSITION OF PATIENTS

This section describes patient disposition for both patient study status and the patient analysis populations.

Screened patients are defined as all patients who have signed the informed consent.

Randomized patients consist of all patients with a signed informed consent form who have had a treatment kit number allocated and recorded in the IRT database, regardless of whether the treatment kit was used or not.

For patient study status, the total number of patients in each of the following categories will be presented in the CSR using a flowchart diagram or summary tables:

- Screened patients.
- Run in patients: patients who had a run-in record in IRT.
- Screen failure patients (including failures during run-in) and reasons for screen failure.
- Nonrandomized but treated patients.
- Randomized patients.

- Randomized but not treated patients.
- Randomized and treated patients.
- Patients who have completed the 26-week double-blind core treatment period (see Section 2.5.4) as per protocol.
- Patients did not complete the 26-week double-blind core treatment period (see Section 2.5.4) as per protocol and the reasons for permanent treatment discontinuation.
- Patients who have completed the 79-week entire treatment period as per protocol (double-blind core treatment period and extension treatment period).
- Patients who did not complete the 79-week entire treatment period as per protocol, and the reasons for permanent treatment discontinuation.
- Patients who have completed the study as per protocol.
- Patients who did not complete the study as per protocol and the reasons for study discontinuation.
- Patients' end of study status (completed, not completed) and corresponding end of entire treatment status (completed, not completed).
- Status at last study contact.

For screened, run in, screen failure, and nonrandomized but treated patients, percentages will be calculated using the number of screened patients as the denominator. All other categories of patients will be presented by treatment group and the percentages will be calculated using the number of randomized patients within each treatment group as the denominator. Reasons for treatment discontinuation will be supplied in tables giving numbers and percentages by treatment group. Patients prematurely discontinued from treatment and/or study, along with reasons for discontinuation, will also be listed.

A summary of the distribution of patients by country and center will also be provided (overall number of patients screened, run-in, randomized, and treated, as well as number of patients randomized, discontinued from study treatment, and discontinued from study for each treatment group).

Patients treated but not randomized, patients randomized but not treated and patients randomized but not treated as randomized will be identified and described in separate listings. The patients of the third category (randomized and not treated as randomized) will be part of efficacy and safety analyses (Section 2.3). Patients randomized but not treated will be included in efficacy analysis. Safety data of patients treated but not randomized will be reported separately.

The randomization strata [HbA1c at Screening ( $\leq$ 8.5%, >8.5%), Metformin use at screening (Yes, No), and mean SBP at Screening (<130,  $\geq$ 130 mmHg)] assigned by IRT will be summarized. The percentages will be calculated using the number of randomized patients as the denominator. The discrepancy between the strata assigned by IRT and the information reported on e-CRF will be listed for all randomized patients.

Kaplan-Meier (KM) plots of the cumulative incidence of double-blind IMP discontinuations due to any reason and due to AE will be provided for the entire 79-week double-blind treatment period separately. A listing of these patients, along with the reason for discontinuation of treatment, study completion status and the reason for discontinuation study, will be provided.

All important deviations including randomization and drug-dispensing irregularities will be summarized in tables giving numbers and percentages of deviations by randomized treatment group.

Additionally, the analysis populations for safety, efficacy, and pharmacokinetics defined in Section 2.3 will be summarized in a table by number of patients in the randomized population.

- Efficacy population: intent-to-treat (ITT) population.
- Safety population.
- PK population.

## 2.2.1 Randomization and drug dispensing irregularities

Randomization and drug-dispensing irregularities occur whenever:

- A randomization is not in accordance with the protocol-defined randomization method, such as a) an ineligible patient is randomized, b) a patient is randomized based on an incorrect stratum, c) a patient is randomized twice, or d) in a dynamic randomization scheme the treatment assignment is, in fact, not random, due to a computer program error.
  - OR
- 3. A patient is dispensed an IMP kit not allocated by the protocol-defined randomization, such as a) a patient at any time in the study is dispensed a different treatment kit than as randomized (which may or may not contain the correct-as-randomized IMP), or b) a nonrandomized patient is treated with IMP reserved for randomized patients.

Randomization and drug-dispensing irregularities will be monitored throughout the study and reviewed on an ongoing basis.

All randomization and drug-dispensing irregularities will be documented in the CSR. If the number of irregularities is large enough to make a tabular summary useful, the irregularities will be categorized and summarized among randomized patients (number and percentages). Nonrandomized, treated patients will be described separately. Listings with additional, relevant details will be provided in appendices.

Randomization and drug-dispensing irregularities to be prospectively identified include but are not limited to:

#### Randomization and drug allocation irregularities

Kit dispensation without IRT transaction

Erroneous kit dispensation

Kit not available

Randomization by error

Patient randomized twice

Stratification error

Patient switched to another site

#### 2.3 ANALYSIS POPULATIONS

Patients treated without being randomized will not be considered randomized and will not be included in any efficacy population.

The randomized population includes any patient who has been allocated to a randomized treatment regardless of whether the treatment kit was used.

For any patient randomized more than once, only the data associated with the first randomization will be used in any analysis population. The safety experience associated with any later randomization will be assessed separately.

The safety experience of patients treated and not randomized will be reported separately, and these patients will not be in the safety population.

#### 2.3.1 Efficacy populations

Efficacy analyses will be based on the treatment group allocated by the IRT according to the randomization schedule at randomization visit (as randomized), irrespective of the treatment actually received.

#### 2.3.1.1 Intent-to-treat population

Efficacy analyses will be based on the ITT population, defined as all randomized patients, irrespective of compliance with the study protocol and procedures. Patients will be analyzed for efficacy according to the treatment group to which they are randomized.

## 2.3.2 Safety population

Safety analyses will be based on the safety population, defined as all randomized patients who receive at least one dose or part of a dose of double-blind IMP(regardless of the amount of treatment administered). Patients will be analyzed according to the treatment actually received.

#### In addition:

- Nonrandomized but treated patients will not be part of the safety population; however, their safety data will be presented separately.
- Randomized patients for whom it is unclear whether they took the IMP will be included in the safety population as randomized.
- When a patient is exposed to both placebo and sotagliflozin, the patient will be analyzed in the sotagliflozin 400 mg group.
- Randomized patients will be excluded from the safety population only if there is
  documented evidence (ie, all study dates recorded as no medication taken) that patients
  have not taken the study treatment. If a patient is dispensed double-blind IMP and is lost to
  follow-up without any documented evidence, the patient will be considered exposed.

### 2.3.3 Pharmacokinetic population

For PK analyses, the PK population is defined as all safety patients who contribute with at least 1 valid plasma concentration of sotagliflozin or its 3-O-glucuronide metabolite. The PK data will be analyzed according to the treatment actually received (See Section 2.3.2).

#### 2.4 STATISTICAL METHODS

### 2.4.1 Demographics and baseline characteristics

Continuous data will be summarized using the number of observations available, mean, SD, median, minimum, and maximum for each treatment group. Categorical and ordinal data will be summarized using the count and percentage of patients in each treatment group.

Parameters will be summarized based on the randomized population analyzed in the treatment group to which they were randomized. Analyses for the safety population will be included in the appendices if the size of the safety population is different (>10%) from the size of that in the primary analysis population (ie, randomized patients) for any treatment group.

Parameters described in Section 2.1.1 will be summarized by treatment group and overall (pooled across treatment groups) using descriptive statistics.

P-values on the treatment difference for the demographic and baseline characteristic data will not be calculated.

In general, no specific description of the safety parameters will be provided at baseline. If relevant, the baseline values will be described along with each safety analysis.

In general, no specific description of the efficacy parameters will be provided at baseline. If relevant, the baseline values will be described along with each efficacy analysis.

#### 2.4.2 Prior or concomitant medications

The prior, concomitant and posttreatment medications will be presented in the randomized population for each treatment group (and overall for the summary of prior medications), using counts and percentages. No statistical test for the between-group difference will be performed.

Medications will be summarized by treatment group according to the WHO-DD dictionary, considering the first digit of the anatomical therapeutic chemical (ATC) class (anatomic category) and the first 3 digits of the ATC class (therapeutic category). A given medication may be classified in more than 1 ATC class. All ATC codes corresponding to a medication will be summarized, and a patient will be counted once within each ATC category (anatomic or therapeutic) linked to the medication. Therefore a patient may be counted several times for the same medication.

Prior medications will be presented by anatomic and therapeutic categories and sorted by decreasing frequency of ATC based on the overall incidence across treatment groups. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

Concomitant and posttreatment medications will be presented by anatomic and therapeutic categories and sorted by decreasing frequency in the sotagliflozin 400 mg group. In case of equal frequency regarding ATCs (anatomic or therapeutic categories), alphabetical order will be used.

## 2.4.3 Extent of investigational medicinal product exposure and compliance

The extent of IMP exposure and compliance will be assessed and summarized by actual treatment within the safety population (Section 2.3.2).

## 2.4.3.1 Extent of investigational medicinal product exposure

The extent of IMP exposure will be assessed by the duration of IMP exposure.

Duration of IMP exposure is defined as last dose date of double-blind IMP – first dose date of double-blind IMP + 1 day, regardless of unplanned intermittent discontinuations (see Section 2.5.3 for calculation in case of missing or incomplete data). Duration of IMP exposure will be summarized descriptively as a quantitative variable (number of patients exposed, mean, SD, median, minimum, and maximum). In addition, duration of treatment exposure will also be summarized categorically by numbers and percentages for each of the following categories and cumulatively according to these categories:

- 1 to 28 days,
- 29 to 56 days,
- 57 to 84 days,
- 85 to 126 days,
- 127 to 182 days,

- 183 to 364 days,
- 365 to 551 days,
- >551 days.

Additionally, the cumulative duration of treatment exposure will be provided, defined as the sum of the duration of treatment exposure for all patients, and will be expressed in patient years.

Number and percentage of patients by final dose at the end of the treatment will also be presented by each treatment group.

## 2.4.3.2 Compliance

A given administration will be considered noncompliant if the patient did not take the planned dose of treatment as required by the protocol. No imputation will be made for patients with missing or incomplete data.

Percentage of compliance for a patient will be defined as the number of days that the patient was compliant divided by the total number of days that the patient was planned to take during the treatment epoch defined in Section 2.1.4 (ie, from the first date to the last date of double-blind IMP administration).

Above-planned dosing percentage for a patient will be defined as the number of days that the patient took a higher dose than planned divided by the total number of days that the patient was planned to take during the treatment epoch.

Under-planned dosing percentage for a patient will be defined as the number of days that the patient took a lower dose than planned divided by the total number of days that the patient was planned to take during the treatment epoch.

Treatment compliance, above-planned, and under-planned dosing percentages will be summarized descriptively as quantitative variables (number, mean, SD, median, minimum, and maximum). The percentage of patients whose compliance is <80% will be summarized. In addition, numbers and percentages of patients with at least 1 day above-planned dose administration will be provided, as well as numbers and percentages of patients with (0, 20%], and >20% of days under-planned dose administrations.

Cases of overdose (see study protocol for further details) will constitute AEs/SAEs and be analyzed as such. More generally, dosing irregularities will be listed in Section 2.2.1.

## 2.4.4 Analyses of efficacy endpoints

Efficacy analyses will be performed on the ITT population using the efficacy assessments collected during the study, including those obtained after IMP discontinuation or introduction of rescue therapy, unless otherwise specified.

Statistical testing will be performed for primary endpoint and some secondary endpoints at Week 26 (or Week 12 for SBP) as specified in following subsections. All efficacy variables after Week 26 will only be summarized by descriptive statistics without formal statistical testing.

Missing data for efficacy analyses is identified through steps described in Section 2.5.4.

## 2.4.4.1 Analysis of primary efficacy endpoint

The statistical test will be two-sided tests at a nominal 5% significance level.

## Primary analysis

The primary efficacy endpoint of change in HbA1c from baseline to Week 26 will be analyzed by an Analysis of Covariance (ANCOVA) model using HbA1c values measured at baseline and Week 26 (observed or imputed). The missing data at endpoint will be imputed by multiple imputation [MI]) methods as detailed below. To be concise, the following texts related to imputation are generalized to accommodate primary as well as continuous secondary efficacy endpoints.

Missing endpoint data at Week 26 (or Week 12 for SBP) visit will be imputed using a model built separately in each treatment group and estimated from the patients in the same treatment group who prematurely discontinue the IMP before the Week 26 (or Week 12 for SBP) visit but have the measurement for the endpoint (ie, retrieved dropouts). The imputation model will include the randomization strata and the corresponding baseline value. In cases of non-convergence during the imputations, the offending stratum will be identified and then will be dropped from the model. Considering that the number of retrieved dropout patients in each treatment group is expected to be small, a simple imputation model based on regression will be used with baseline measurement included as the predictor. This will serve as the primary method of imputation for missing data should sampling criteria be satisfied (see below).

An alternative (back-up) imputation method will be used if the number of patients who prematurely discontinue the IMP before the Week 26 (or Week 12 for SBP) visit but have the measurement for the endpoint is < 5 in any treatment groups (ie, an insufficient number of retrieved dropouts to support the imputation method described above). This criterion will be assessed for each primary and continuous secondary efficacy endpoint.

In the back-up imputation method, missing post-baseline endpoint values at Week 26 (or Week 12 for SBP) will be imputed by the washout Multiple Imputation (MI) method under the missing not at random (MNAR) framework.

Missing endpoint data at the Week 26 (or Week 12 for SBP) in all treatment groups (sotagliflozin 400 mg and placebo) are imputed from a model estimated from patients in the placebo group who have the endpoint data available.

For patients in the sotagliflozin 400 mg group with missing data at Week 26 (or Week 12 for SBP), their missing values will be imputed using observed baseline and the observed primary endpoint data from placebo completers; no intermittent values from either placebo or the active treatment groups will be used.
For placebo patients, missing data will be imputed based on the placebo group data. Intermittent observed values will be used while imputing missing values at Week 26 (or Week 12 for SBP). In cases that a non-monotone missing data pattern occurs at the intermediate visits, these data points will be first imputed in the placebo group using the Markov Chain Monte Carlo (MCMC) option in PROC MI to achieve a monotone missing pattern for all placebo patients. The Week 26 (or Week 12 for SBP) endpoint values will be subsequently imputed from the multiple copies of the original dataset where each copy will have a monotone missing pattern.

The imputation models for the washout MI method will include the randomization strata and the corresponding baseline value. Missing data will be imputed using the regression method.

In cases of non-convergence during the imputations, especially for the MCMC application in the placebo non-monotone datasets, graphical measures (eg, trace and autocorrelation plots) will be used to identify the offending variable and once detected, that variable(s) will be dropped from the model and the imputations will be re-run. These re-run models will use the same seed number and number of imputations as used in the original models.

Using either imputation method, missing endpoint data will be imputed 2000 times to generate multiple data sets with complete data. Other details of the imputation procedures such as the seed number and sort ordering are specified in the SAS programs. The HbA1c change from baseline to Week 26 (or Week 12 for SBP) will be derived from observed and imputed HbA1c values at Week 26 (or Week 12 for SBP).

Each of the completed datasets after the imputation will be analyzed using the Analysis of Covariance (ANCOVA) model with treatment groups (sotagliflozin 400 mg, placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg, ≥130 mmHg), and country as fixed factors, and baseline value of the efficacy endpoint as a covariate.

Results from each analysis will be combined using Rubin's formula, to provide the adjusted mean change in HbA1c from baseline to Week 26 (or Week 12 for SBP) for each treatment group, as well as the between-group difference (comparing sotagliflozin 400 mg versus placebo) and its associated 95% confidence interval (CI).

#### Sensitivity analyses

Tipping point analysis based on the same MI method as applied to the primary analysis will be performed to examine the robustness of the results from the primary analysis. Patients who were randomized to sotagliflozin 400 mg group and had no HbA1c data at Week 26 will be given a penalty. The penalty will be gradually increased to evaluate at which level the conclusion of the analyses in terms of statistical significance is changed. The tipping point is the penalty level, at which the magnitude of efficacy reduction in patients without HbA1c data at Week 26 creates a shift in the treatment effect of sotagliflozin 400 mg from being statistically significantly better than placebo to a non-statistically significant effect. LS mean difference between sotagliflozin 400 mg and placebo and its associated p-value will be provided for each penalty level. The steps to perform the tipping point analysis are as follows:

1. Missing data will be imputed using the same MI method as applied to the primary analysis..

- 2. The imputed HbA1c value at Week 26 in the sotagliflozin 400 mg group will be penalized by adding a penalty  $\delta$  (eg,  $\delta$  = 0.1%) in each complete dataset..
- 3. Change from baseline at Week 26 in HbA1c will be analyzed using the same ANCOVA model as specified in the primary analysis in each complete dataset..
- 4. Results will be combined across complete datasets using Rubin's formula...
- 5. Steps 2 to 4 will be repeated with incremental penalty at δ (ie, δ, 2δ, 3δ, .....) until the p-value for treatment effect of sotagliflozin 400 mg compared to placebo estimated in Step 4 is >0.05.

The tipping point analysis will be performed on the ITT population. The tipping point analysis will be performed for the primary variable only if that variable (change from baseline to Week 26 in HbA1c comparing sotagliflozin 400 mg vs. placebo) is statistical significant at  $\alpha = 0.05$  (2-sided).

In addition to the tipping point analyses, if the retrieved dropout imputation is applied to the primary analysis, the analysis based on the washout imputation method (ie, the backup imputation method) will be presented as a sensitivity analysis.

Patients in this study have undergone sampling for plasma levels of sotagliflozin and its main active metabolite in order to perform population PK analysis. Patients may be identified as those who have no detectable levels of active study drug or metabolite in their samples (ie, Below Limit of Quantification or BLOQ). When sample analysis has been completed and the study has been unblinded, explanations for some of these patients may be found: known non-compliance or sampling occurring after treatment had been discontinued. In other cases, drug intake history relative to the randomization assignment may not be fully explained. The ITT-based analyses specified in this document provides for a conservative assessment of the efficacy data should patients have been subjected to these unexplained non-compliance findings or PK 'anomalies'. To provide a broader perspective on the impact of these apparent errors in compliance, additional sensitivity analyses of the primary efficacy endpoint and continuous efficacy endpoints may be conducted. The need to perform such analyses, their specifics, and results will be provided in the Clinical Study Report (CSR), if applicable. The analysis methods applied to the patient subpopulations defined by the occurrence of the PK anomalies (eg, exclusion of patients with PK anomalies from the ITT dataset) will include the ANCOVA model using the retrieved dropout and/or washout MI methods previously specified in this section.

#### Assessment of treatment effect by subgroup

Descriptive analyses will be performed on the primary endpoint to summarize the treatment effects across subgroups defined by the following Baseline or Screening factors:

- Race (White, Black or African American, Asian, Other) (any race groups with fewer than 5 patients may be combined with "Other" category as appropriate).
- Ethnicity (Hispanic, Not Hispanic).
- Age group (<50, ≥50 to <65, ≥65 years) (any category with fewer than 5 patients may be combined with another category as appropriate).

- Gender (Male, Female).
- Baseline BMI level ( $<30, \ge 30 \text{ kg/m}^2$ ).
- Baseline HbA1c (<8.5%, >8.5%).
- Metformin use at Screening (Yes, No).
- Baseline mean SBP (<130 mmHg, ≥130 mmHg).</li>
- Baseline eGFR (≥30 to <60 mL/min/1.73m<sup>2</sup> [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m<sup>2</sup> [Mild decrease in GFR], and ≥90 mL/min/1.73m<sup>2</sup> [Normal]).
- Duration of diabetes (<10, ≥10 years).</li>
- Country.

The treatment effects (sotagliflozin 400 mg versus placebo) across the subgroups defined for each of these factors will be estimated for the change from Baseline to Week 26 in HbA1c in the ITT population , and using the same MI method as applied to the primary analysis. The ANCOVA model will include treatment groups (sotagliflozin 400 mg, placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg, ≥130 mmHg), subgroup factor, treatment-by-subgroup factor, and country as fixed factors and baseline HbA1c values as a covariate. The adjusted estimates of treatment mean differences (sotagliflozin 400 mg versus placebo) with standard error (SE) and 95% CIs will be provided as appropriate across the subgroups. A graphical presentation of the results (ie, forest plot) will also be provided.

In the case that the subgroup factor is identical or similar to a randomization strata factor (eg, baseline HbA1c, metformin use at screening, or baseline mean SBP category), only the subgroup factor (as a single factor or an interaction term) will be included in the model in order to avoid the issue of collinearity in the analysis. The corresponding strata factor will not be included in the model.

## Summary statistics at scheduled visits

Summary statistics (for screening value, baseline value, observed post-baseline value and its changes from baseline) at scheduled visits will be provided for each treatment group. The summary will include the number of observations, mean, SD, SE, minimum, median, and maximum. Graphical presentations will also be used to examine trends over time using mean values (±SE) and mean changes from baseline (±SE) at each of the scheduled visits.

Similar presentations will be provided excluding measurements after rescue therapy during the entire 79-week double-blind treatment period.

#### 2.4.4.2 Analyses of secondary efficacy endpoints

For continuous secondary efficacy parameters with missing data at baseline, missing baseline data will be imputed using MI under the missing at random (MAR) assumption. Missing data at baseline will be imputed using regression method that includes randomization stratum of HbA1c

( $\leq$ 8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg,  $\geq$ 130 mmHg), and baseline value in the imputation model..

Each continuous secondary efficacy endpoint (Section 2.1.3.2) will be analyzed using a similar ANCOVA model including the measurements at baseline and endpoint (observed or imputed). The missing data at endpoint will be imputed by the retrieved dropouts if there are at least 5 patients in each study treatment group who discontinued but have the endpoint. Otherwise, the washout imputation method will be used according to the criterion described in Section 2.4.4.1. After the imputation, each of the complete datasets will be analyzed by an ANCOVA model.

The ANCOVA model will include treatment groups (sotagliflozin 400 mg, placebo), randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), randomization stratum of SBP (<130 mmHg, ≥130 mmHg), and country as fixed effects, and the corresponding baseline secondary endpoint value as a covariate. For the analysis of SBP in patients with baseline SBP ≥130 mmHg, the randomization stratum of SBP will not be included in the ANCOVA model. Results from each complete dataset will be combined using Rubin's formula to provide the adjusted mean change from Baseline to Week 26 (or Week 12 for SBP) for each treatment group, as well as the between-group difference (comparing sotagliflozin 400 mg versus placebo) and the 95% CI for the difference.

For all continuous secondary endpoints, summary statistics at scheduled visits will be provided for each treatment group. The summary will include the number of observations, mean, SD, SE, minimum, median, and maximum. Graphical presentations will also be used to examine trends over time using mean values ( $\pm$ SE) and mean changes from baseline ( $\pm$ SE) at each of the scheduled visits. In addition, SBP will be summarized descriptively at each visit for those patients with baseline SBP  $\geq$ 140 mmHg.

The categorical secondary efficacy variables of HbA1c <6.5%, <7% at Week 26 will be analyzed respectively using a Cochran-Mantel-Haenszel (CMH) method stratified by randomization stratum of HbA1c (≤8.5%, >8.5%), randomization stratum of metformin use at Screening (Yes, No), and randomization stratum of SBP (<130 mmHg, ≥130 mmHg). The proportion in each treatment group will be provided, as well as the difference of proportions between sotagliflozin 400 mg and placebo with the associated 2-sided 95% CI. For HbA1c responders at Week 26 (<6.5%, <7% respectively), all values at Week 26 will be used to determine whether a patient is a responder or not, even if they are measured after IMP discontinuation or rescue medication use. Patients who have no HbA1c measurement at Week 26 will be treated as non-responders. Summary tables and graphs will also be provided by treatment group at scheduled visits.

For between-group comparison, a sensitivity analysis will be performed respectively for HbA1c <6.5% responder analysis by excluding patients whose HbA1c values at baseline are <6.5%, and for HbA1c <7% responder analysis by excluding patients whose HbA1c values at baseline are <7% using the same CMH test mentioned above. Similarly, by-visit summary may also be provided excluding those patients.

## 2.4.4.3 Analyses of other efficacy endpoints

The analysis of other endpoints (see Section 2.1.3) will be descriptive with no formal testing. Summary statistics at scheduled visits based on observed value will be provided by each treatment group. Graphical presentations will also be used to illustrate trends over time as appropriate.

The number (%) of patients who used rescue therapy will be summarized by treatment group during the core (see Section 2.5.4) and the entire double-blind treatment periods. A KM curve for the time to first rescue therapy will be provided by treatment group. A list of patients who used rescue therapy will also be provided (see Section 2.5.4).

## 2.4.4.4 Multiplicity issues

To control the family-wise type I error, a fixed sequence testing procedure will be applied.

Once the primary hypothesis (superiority of the change from Baseline to Week 26 in HbA1c comparing sotagliflozin 400 mg versus placebo) is statistically significant for the primary efficacy endpoint at  $\alpha = 0.05$  (2-sided), the following secondary hypothesis based on change from Baseline scores will be tested in the following prioritized order:

- 1. Change from Baseline to Week 26 in FPG.
- 2. Change from Baseline to Week 26 in body weight.
- 3. Change from Baseline to Week 12 in SBP for patients with baseline SBP ≥130 mmHg.
- 4. Change from Baseline to Week 12 in SBP for all patients.
- 5. Proportion of patients with HbA1c <7.0% at Week 26.

If any hypothesis is found to be not statistically significant, the testing procedure will be stopped and the following hypotheses will not be tested.

No multiplicity adjustment will be made on other secondary efficacy variables than mentioned above.

### 2.4.5 Analyses of safety data

The summary of safety results will be presented by treatment group.

Safety endpoints are presented in Section 2.1.4. The summary of safety results will be presented by treatment group. The safety data will be summarized for the 26-week core treatment period and the 79-week entire treatment period separately, unless otherwise specified.

The "observation period" defined in Section 2.1.4 is applicable in all safety analyses for the classification of AEs, determination of treatment-emergent PCSA values and the last on-treatment value for the laboratory, vital sign and ECG.

#### General common rules

All safety analyses will be performed on the safety population as defined in Section 2.3.2, unless otherwise specified, using the following common rules:

- Safety data in patients who do not belong to the safety population (eg, exposed but not randomized) will be listed separately.
- The baseline value (with the exception of serum creatinine and eGFR) is defined as the
  last available value before the first dose of double-blind IMP, with the exception of
  creatinine and eGFR, where the baseline value is defined as the average of all values
  before the first dose of double-blind IMP.
- PCSA values are defined as abnormal values considered medically important by the Sponsor according to predefined criteria/thresholds based on literature review and defined by the Sponsor for clinical laboratory tests, vital signs, and ECG (Appendix A).
- PCSA criteria will determine which patients had at least 1 PCSA during the TEAE period, taking into account all evaluations performed during the TEAE period, including nonscheduled or repeated evaluations. The number of all such patients will be the numerator for the treatment-emergent PCSA percentage.
- The treatment-emergent PCSA denominator by group for a given parameter will be based on the number of patients assessed for that given parameter during the TEAE period by treatment group in the safety population.
- For laboratory parameters cited in the protocol as efficacy endpoints (including HbA1c and plasma glucose etc.), PCSA summaries will not be provided. These parameters will be summarized in efficacy Section 2.4.4. For creatinine and eGFR, PCSA summaries will be presented in safety Section 2.4.5 while descriptive summaries in efficacy Section 2.4.4.
- For quantitative safety parameters based on central laboratory/reading measurements, descriptive statistics will be used to summarize results and change from baseline values by visit and treatment group for the 79-week entire treatment period only. Summaries will include the last on-treatment value. The last on-treatment value is commonly defined as the value collected at the same day/time of the last administration of IMP for the 79-week entire treatment period. If this value is missing, this last on-treatment value will be the closest value prior to the last administration of IMP during the 79-week entire treatment period.
- The analysis of the safety variables will be essentially descriptive and no statistical testing is planned. Relative risks versus placebo and their 95% CIs may be provided, if relevant.
- Selected safety analyses will be summarized by age, gender, racial subgroups, and other pertinent subgroups (see details in Section 2.4.5.1 and Section 2.4.5.2).

# 2.4.5.1 Analyses of hypoglycemia

Analyses of hypoglycemia will be performed on the TEAE periods as defined in Section 2.1.4. Hypoglycemia will be classified as severe hypoglycemia, documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia or relative hypoglycemia Section 2.1.4.1.

The number (%) of patients with any hypoglycemia, severe hypoglycemia, and documented symptomatic hypoglycemia will be summarized respectively by treatment group during the TEAE period, as well as the incidence rate in patient years. Two types of incidence rates will be presented: the number of patients with at least 1 event per 100 patient years (calculated as the number of patients with at least 1 event / total exposure in 100 patient years), and the number of events per 100 patient-years [calculated as the total number of events / (total exposure in 100 patient-years)]. Note: here exposure (in days) is duration of TEAE period, ie, duration of IMP treatment in days +1 (Section 2.1.4).

The summary of frequency and incidence rate in patient years for severe hypoglycemia or documented symptomatic hypoglycemia will be provided as appropriate by gender (Male, Female), age group ( $<50, \ge 50$  to  $<65, \ge 65$  years),race (White, Black or African American, Asian, Other) and Metformin use at Screening (Yes, No).

A KM curve will also be provided by treatment group for the time to first severe hypoglycemia or documented symptomatic hypoglycemia during the TEAE period for the 79-week entire treatment period only.

Documented symptomatic hypoglycemia maybe presented by  $\leq$ 3.9 mmol/L ( $\leq$ 70 mg/dL) and  $\leq$ 3.0 mmol/L ( $\leq$ 54 mg/dL) respectively, as appropriate.

A listing of patients for all events reported on the dedicated e-CRF "Hypoglycemic event information" page will be provided with each category flagged (ie, severe hypoglycemia, documented symptomatic hypoglycemia, asymptomatic hypoglycemia, probable symptomatic hypoglycemia and relative hypoglycemia).

# 2.4.5.2 Analyses of adverse events

## Generalities

The primary focus of adverse event reporting will be on TEAEs. Pretreatment and posttreatment AEs will be described separately.

If an AE date/time of onset (occurrence, worsening, or becoming serious) is incomplete, an imputation algorithm will be used to classify the adverse event as pretreatment, treatment-emergent, or posttreatment. The algorithm for imputing date/time of onset will be conservative and will classify an AE as treatment emergent unless there is definitive information to determine it is pretreatment or posttreatment. Details on classification of AEs with missing or partial onset dates are provided in Section 2.5.3.

Adverse event incidence tables will be presented by SOC, HLGT, HLT, and PT, sorted by the internationally agreed order for SOCs and alphabetic order for HLGT, HLT and PT within a SOC, the number (n) and percentage (%) of patients experiencing an adverse event. Multiple occurrences of the same event in the same patient will be counted only once in the tables within a treatment phase. The denominator for computation of percentages is the safety population within each treatment group.

Sorting within tables ensures the same presentation for the set of all AEs within the observation period (pretreatment, treatment-emergent, and posttreatment). For that purpose, the table of all TEAEs presented by primary SOC and PT (sorted by the internationally agreed SOC order and decreasing frequency of PTs within SOCs in the sotagliflozin 400 mg group) will define the presentation order for all other similar tables unless otherwise specified. In case of equal frequency regarding PTs, alphabetical order will be used.

### Analysis of all TEAEs

The following TEAE summaries will be generated during the 26-week core and the 79-week entire treatment periods respectively in the safety population.

- Overview of TEAEs, summarizing number (%) of patients with any
  - TEAE,
  - Serious TEAE,
  - TEAE leading to death,
  - TEAE leading to permanent treatment discontinuation.
- All TEAEs by primary SOC, showing number (%) of patients with at least 1 TEAE, sorted by internationally agreed order of primary SOC.
- All TEAEs by primary SOC, HLGT, HLT, and PT, showing number (%) of patients with at least 1 TEAE sorted by the SOC internationally agreed order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.
- Number (%) of patients experiencing TEAE(s) presented by PT, sorted by decreasing incidence of PT in the sotagliflozin 400mg group.
- All TEAEs by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE, sorted by the internationally agreed SOC order and by decreasing incidence of PTs within each SOC in the sotagliflozin 400mg group. This sorting order will be applied to all other similar tables, unless otherwise specified.
- All TEAEs regardless of relationship and related to IMP by primary SOC, HLGT, HLT and PT, showing the number (%) of patients with at least 1 TEAE, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.
- All TEAEs by maximal severity, presented by primary SOC and PT, showing the number (%) of patients with at least 1 TEAE by severity (ie, mild, moderate, or severe), sorted by the sorting order defined above.
- Common TEAEs (PTs with an incidence ≥2% in any treatment group) by primary SOC, HLGT, HLT, and PT, sorted by internationally agreed order of SOCs. The other levels (HLGT, HLT, PT) will be presented in alphabetic order.

- Common TEAEs (PTs with an incidence ≥2% in any treatment group) will be provided as appropriate by primary SOC, and PT and by demographic factors including gender (Male, Female), age group (<50, ≥50 to <65, ≥65 years of age), race (White, Black or African American, Asian, other), baseline SBP category (<130 mmHg, ≥130 mmHg), Metformin use at Screening (Yes, No), and baseline eGFR category (≥30 to <60 mL/min/1.73m² [Moderate decrease in GFR], ≥60 to <90 mL/min/1.73m² [Mild decrease in GFR], and ≥90 mL/min/1.73m² [Normal]). SOC will be sorted by internationally agreed order and the PT by decreasing incidence within each SOC in the sotagliflozin 400 mg group, as described above.
- TEAEs (PTs with an incidence ≥5% in any treatment group) by primary SOC, HLGT, HLT, and PT, sorted by internationally agreed order of SOCs. The other levels (HLGT, HLT, PT) will be presented in alphabetic order.

## Analysis of all treatment emergent SAE(s)

- All treatment-emergent SAEs by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients with at least 1 serious TEAE, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order
- All treatment-emergent SAEs regardless of relationship and related to IMP, by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients with at least 1 treatment-emergent SAE, sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.

## Analysis of all TEAE(s) leading to treatment discontinuation

 All TEAE leading to treatment discontinuation, by primary SOC, HLGT, HLT, and PT, showing the number (%) of patients sorted by the internationally agreed SOC order. The other levels (HLGT, HLT, PT) will be presented in alphabetical order.

#### Analysis of AESI

The summaries of AESI will be presented for the 79-week entire treatment period only in the safety population.

Pregnancy and overdose will be included in overall AE summaries if any are reported. ALT increase >3 x ULN is included in laboratory PCSA summary if any.

The number (%) of patients with an AESI will be summarized by PT and by treatment group during the 79-week entire treatment period only. Corresponding listings will be provided as appropriately.

### Analysis of EOSI

The summaries of EOSI will be presented for the 79-week entire treatment period only in the safety population.

CV events, bone fracture and DKA

For EOSIs that are adjudicated (ie, deaths, myocardial infarction, stroke, and unstable angina requiring hospitalization, heart failure requiring hospitalization, bone fracture, and diabetic ketoacidosis), the number (%) of patients with an EOSI positively adjudicated by CEC will be summarized by treatment group. All EOSIs sent for adjudication and/or reported by the investigators in the specific AE forms will be listed along with the adjudication outcome.

#### Renal events

For the EOSI renal events where selected events are adjudicated, the number (%) of patients with any renal events identified in Table 3 in Section 2.1.4.2 will be summarized by treatment group.

The following renal events will be listed along with the adjudication outcome if applicable, including events,

- i. recorded in e-CRF "GFR decrease",
- ii. recorded in e-CRF "Renal Event Dialysis",
- iii. identified as "Renal transplant" in e-CRF "Other procedure",

Renal death will be part of all deaths specified above.

### Other EOSIs

For EOSIs that are not adjudicated, the number (%) of patients with at least one event will be summarized by treatment group and by PT (as identified in Table 3 in Section 2.1.4.2).

Severe hypoglycemia will be included in the summary of hypoglycemia (See Section 2.5.1).

AE leading to an amputation is described in the section below.

#### Analysis of Amputation

The number (%) of patients with amputation will be summarized by treatment group and by PT and LLT during the study (ie, regardless of on- or post-treatment). Amputation is a procedure recorded in e-CRF "Other Procedures related to Amputation". Patients who had a procedure related to amputation will be listed.

The number (%) of patients with an "AE leading to an amputation" will be summarized by treatment group and by PT. The "AE leading to an amputation" is determined by the AE identifier recorded in e-CRF "Other Procedures related to Amputation" when "AE correction" is chosen as the reason for the amputation procedure.

In addition, the number (%) of patients with an "AE potentially leading to an amputation" will be summarized by treatment group and by PT (as identified in Table 3 in Section 2.1.4.2; these PTs in Table 3 were requested by the European Medicines Agency/ Pharmacovigilance Risk Assessment Committee[EMA/PRAC] Assessment Report 9 February 2017). Associated list will be provided as well, with patients who had an amputation procedure flagged. "AE potentially leading to an amputation" represents the condition that may potentially lead to the amputation procedure, but not in all cases an amputation has occurred (as per the EMA/PRAC request).

## Analysis of pretreatment and posttreatment AEs

- All pretreatment AEs by primary SOC and PT, showing the number (%) of patients with at least 1 pretreatment AE, sorted by the internationally agreed SOC order and decreasing incidence of PTs within each SOC in the sotagliflozin 400mg group.
- All posttreatment AEs by primary SOC and PT, showing the number (%) of patients with at least 1 posttreatment AE, sorted by the internationally agreed SOC order and decreasing incidence of PTs within each SOC in the sotagliflozin 400mg group.

### **Listings**

Supportive AE listings will be provided for all AEs, SAEs, and death, AEs leading to treatment discontinuation and/or death, and EOSI as appropriate. Listing of all AEs, SAEs and AEs leading to treatment discontinuation and/or death will include at least the following information, sorted by treatment, patient identification, and onset date: treatment, patient identification, country, age, gender, race, BMI, primary SOC, PT, reported term, onset date, study day (relative day to the start date of double-blind treatment), AE duration, duration of exposure, intensity, corrective treatment, action taken with IMP, date of treatment discontinuation (if relevant), relationship to IMP or NIMP, outcome, date of death (if any), seriousness, seriousness criteria, and AE status ("E" for a TEAE; and "P" for an on-study post-treatment AE).

#### 2.4.5.3 Deaths

The following summaries of deaths will be generated.

- Number (%) of patients who died by study period (on-study, on-treatment, post-study).
- Deaths in nonrandomized patients or randomized but not treated patients.
- TEAEs leading to death (death as an outcome on the AE e-CRF page as reported by the Investigator) by primary SOC, HLGT, HLT, and PT showing number (%) of patients sorted by internationally agreed SOC order, with HLGT, HLT, and PT presented in alphabetical order within each SOC.

## 2.4.5.4 Analyses of laboratory variables

Laboratory parameters will be grouped and summarized by biological function as described in Section 2.1.4.4.

The summary statistics (including number, mean, median, Q1, Q3, standard deviation, minimum and maximum) of all laboratory variables (central laboratory values and changes from baseline) will be calculated for each applicable visit or study assessment (screening, baseline, each postbaseline time point, last on-treatment value) by treatment group.

The incidence of PCSAs (list provided in Appendix A) at any time during the TEAE period will be summarized for each laboratory test by biological function and treatment group whatever the baseline level and/or according to the following baseline status categories:

Normal/missing.

• Abnormal according to PCSA criterion or criteria.

For parameters for which no PCSA criteria are defined, similar table(s) using the normal range will be provided.

All measurements collected during the TEAE period, including values from unscheduled visits, will be considered for the PCSA summaries. These summaries will include patients in the safety population who have at least 1 assessment performed during the TEAE period. When a PCSA definition involves a change from baseline value, patients must also have a baseline value to be included in the summaries, and when required by the definition of the abnormality, patients must also have available laboratory normal ranges.

A listing of patients with at least 1 post-baseline PCSA (or out of normal range when no PCSA criterion is defined) will be provided and will display the entire patients' profile across time for all parameters belonging to the corresponding biological function. Individual data listings will include the following flags when applicable:

- Baseline values will be flagged "B".
- Normal laboratory ranges, available for most laboratory parameters, will be identified as
  ULN and LLN. Baseline, last on-treatment value, and individual data will be flagged "L"
  if the value is below the LLN and will be flagged "H" if it is above the ULN.
- Laboratory PCSA criteria will be used for the corresponding laboratory parameters.
   Values reaching a PCSA limit will be flagged (+, ++, -, or -- depending upon the direction and level of the abnormality). Flags for WBC and differential counts will be determined using data expressed in international units.

For parameters whose PCSA criteria are multiples of the ULN, the parameter's value will also be expressed as a multiple of the ULN in the individual data provided.

### Drug-induced liver injury

The liver function tests, namely AST, ALT, ALP, and total bilirubin, are used to assess possible drug-induced liver toxicity. The proportion of patients with PCSA values at any postbaseline visit by baseline status will be displayed by treatment group for each parameter. The proportion of patients with PCSA values at any postbaseline visit will also be displayed by duration of exposure for each treatment group (only if a tabulation summary is necessary).

Listing of possible Hy's law cases identified by treatment group (eg, patients with any elevated ALT>3 × ULN, and associated with an increase in bilirubin ≥2 × ULN) with ALT, AST, ALP, total bilirubin, and the following complementary parameters (if available): conjugated bilirubin and prothrombin time/international normalized ratio ,creatine phosphokinase, serum creatinine, complete blood count, anti-HAV IgM, anti-HBc IgM, anti-HCV and HCV RNA, anti-CMV IgM and anti-HEV IgM antibodies, auto-antibodies: anti-nuclear, anti-DNA, anti-smooth muscle, Epstein-Barr virus, herpes viruses, and anti-LKM.

## 2.4.5.5 Analyses of vital sign variables

The summary statistics (including number, mean, median, Q1, Q3, standard deviation, minimum and maximum) of heart rate, temperature and respiratory rate (observed values or mean of observed values, and changes from baseline) will be calculated for each applicable visit or study assessment (baseline, post-baseline time points, last on-treatment value) by treatment group.

The incidence of PCSAs at any time during the TEAE period will be summarized by treatment group for SBP, DBP and HR. All measurements collected during the TEAE period, including values from unscheduled visits, will be considered for the PCSA summaries. The summaries will include patients in the safety population who have at least 1 assessment performed during the TEAE period. When a PCSA definition involves a change from baseline value, patients must also have a baseline value to be included in the summaries.

A listing of patients with at least 1 post-baseline PCSA will be provided and will display the patient's profile over time of all vital sign parameters. Individual data listings will include the following flags:

- Baseline values will be flagged "B".
- Parameter values reaching a PCSA limit will be flagged (+, or depending of the direction).

### 2.4.5.6 Analyses of electrocardiogram variables

Shift tables will be provided to present ECG status according to baseline status (Normal/Missing, Abnormal) for each treatment group during the TEAE period. Supportive listings of patients with abnormal ECG status at any post-baseline visit will be provided.

#### 2.4.5.7 Analyses of physical examination variables

Shift tables will be provided to present physical examination findings by body system according to baseline status (Normal/Missing, Abnormal) for each treatment group during the TEAE period. Supportive listings of patients with abnormal findings at any post-baseline visit will be provided.

## 2.4.6 Analyses of pharmacokinetic variables

Plasma concentrations of sotagliflozin and its 3-O-glucuronide metabolite will be summarized by visit and nominal sampling time (pre-dose at Weeks 4, 18, 26, 52, and 79, and 1 hour 30 minutes post-dose at Week 26 and 79) in the PK population (see Section 2.3.3) in the sotagliflozin 400 mg group, using descriptive statistics such as number, geometric mean, coefficient of variation, median, minimum and maximum. Individual plasma concentrations of sotagliflozin and its 3-O-glucuronide metabolite at nominal sampling times will also be listed.

#### 2.5 DATA HANDLING CONVENTIONS

#### 2.5.1 General conventions

The following formulas will be used for computation of parameters.

#### HbA1c

The formula to convert HbA1c from Diabetes Control and Complications Trial (DCCT) aligned value to International Federation of Clinical Chemistry and Laboratory Medicine (IFCC) standardized value is,

IFCC-HbA1c (mmol/mol) =  $[DCCT-HbA1c (\%) - 2.15] \times 10.929$ .

# Renal function formulas

The estimated GFR (mL/min/1.73 m<sup>2</sup>) will be calculated using the 4 variable Modification of Diet in Renal Disease (MDRD) formula:

Standard unit: eGFR (mL/min/1.73 m<sup>2</sup>) = 175 × [Serum Creatinine ( $\mu$ mol/L)/88.4] <sup>-1.154</sup> × Age (year) <sup>-0.203</sup> × 1.212 (if Black) × 0.742 (if female).

Conventional unit: eGFR (mL/min/1.73 m<sup>2</sup>) =  $175 \times \text{Serum Creatinine (mg/dL)}^{-1.154} \times \text{Age (year)}^{-0.203} \times 1.212 \text{ (if Black)} \times 0.742 \text{ (if Female)}.$ 

# Calculation of LDL-C

When TG is lower than or equal to 4.52 mmol/L (400 mg/dL), LDL-C is calculated using the Friedewald equation as:

- In standard unit (mmol/L), TC HDL-C TG/2.17.
- In conventional unit (mg/dL), TC HDL-C TG/5.

#### 2.5.2 Data handling conventions for secondary efficacy variables

Scheduled measurements (see Section 2.5.4) of continuous efficacy variables collected during the study will be used in the analyses including those obtained after IMP discontinuation or introduction of rescue therapy. Continuous secondary efficacy endpoints will be analyzed with missing values imputed by retrieved dropouts MI method or by the washout MI method according to the criterion described in Section 2.4.4.1.

For the categorical secondary efficacy endpoints, data handling conventions are described in Section 2.4.4.2.

#### 2.5.3 Missing data

For categorical variables, patients with missing data are not included in calculations of percentages unless otherwise specified. When relevant, the number of patients with missing data

is presented.

Derived variables will be considered missing if any of the original variables required to calculate them are missing. For example, if either a baseline assessment or an endpoint assessment is missing for a particular patient, then change from baseline at endpoint will be missing. Depending upon the assessment, analyses may not include all patients in the analysis population, because certain patients in the intended population may have missing data.

## Incomplete date of first administration of double-blind IMP

Date/time of first administration is the first non-missing start date/time of double-blind IMP completed in the e-CRF "First dose IMP" module.

For patients who are randomized and dispensed a double-blind treatment kit but who are lost to follow-up just after Visit 3 (eg. only the treatment kit number is reported in the e-CRF "Exposure - treatment period" module without any dose information), the date of first administration will be imputed using the date of randomization. When a patient is randomized but not exposed, "Not taken" should be ticked in the e-CRF "First dose IMP" module.

## Handling of computation of treatment duration if IMP end of treatment date is missing

For the calculation of the treatment duration, the date of the last dose of double-blind IMP is equal to the date of last administration reported on the e-CRF "Treatment status library" page. If this date is missing, the exposure duration should be left as missing.

The last dose administration should be clearly identified in the e-CRF and should not be approximated by the last returned package date.

## Handling of medication missing/partial dates

No imputation of medication start/end dates or times will be performed. If a medication date or time is missing or partially missing and it cannot be determined whether it was taken prior or concomitantly, it will be considered a prior, concomitant, and post-treatment medication.

### Handling of AE/hypoglycemia with missing or partial date/time of onset

Missing or partial adverse event/hypoglycemia onset dates and times will be imputed so that if the partial adverse event/hypoglycemia onset date/time information does not indicate that the AE/hypoglycemia started prior to treatment or after the treatment-emergent AE, the adverse event/hypoglycemia will be classified as treatment-emergent.

No imputation of adverse event end dates/times will be performed. These data imputations are for categorization purpose only and will not be used in listings. No imputation is planned for date/time of adverse event resolution.

## Handling of AEs/hypoglycemia when date and time of first IMP administration is missing

When the date and time of the first double-blind IMP administration is missing, the day of randomization should be considered as the start date of TEAE period (see Section 2.1.4). The exposure duration should be kept as missing.

## Handling of AEs/hypoglycemia when IMP end of treatment date is missing

For the purpose of defining TEAE period, the date of the last administration of double-blind IMP is equal to the date of the last administration reported on the e-CRF "Treatment Status Library" page. If the date of last administration reported on the e-CRF "Treatment Status Library" page is

- Partially missing, it will be imputed with a date as late as possible before or on the date of last available information on e-CRF "Completion of End of Study/Follow-up".
- Completely missing, it will be imputed with the date of last available information on e-CRF "Completion of End of Study/Follow-up" page.

If the date of last available information on e-CRF "Completion of End of Study/Follow-up" page is:

- Partially missing, it will be imputed with a date as late as possible.
- Completely missing, all adverse events occurred on or after the first administration of double-blind IMP will be considered as TEAEs.

# Handling of missing assessment of relationship of AEs to IMP

If the assessment of the relationship to IMP is missing, the relationship to IMP has to be assumed and the AE considered as such in the frequency tables of possibly related AE, but no imputation should be done at the data level.

## Handling of missing severity/grades of AE

If the severity/grade is missing for 1 of the treatment-emergent occurrences of an AE, the maximal severity on the remaining occurrences will be considered. If the severity is missing for all the occurrences, a "missing" category will be added in the summary table.

#### Handling of potentially clinically significant abnormalities

If a patient has a missing baseline he will be grouped in the category "normal/missing at baseline."

For PCSAs with 2 conditions, one based on a change from baseline value or a normal range and the other on a threshold value, with the first condition being missing, the PCSA will be based only on the second condition.

For a PCSA defined on a threshold and/or a normal range, this PCSA will be derived using this threshold if the normal range is missing; eg, for eosinophils the PCSA is > 0.5 GIGA/L or >ULN if ULN  $\ge 0.5$  GIGA/L. When ULN is missing, the value 0.5 should be used.

Measurements flagged as invalid by the laboratory will not be summarized or taken into account in the computation of PCSA values.

#### Linked AEs that worsened or became serious

An AE that worsened or became serious will have a separate record in the data from the original event record with an AE identification number that links the new record to the original record. An AE that worsened or became serious will be considered a new recurring AE in the summary of recurrent events or in the summary of events by time intervals.

### Handling of missing data for continuous efficacy endpoints

See Section 2.4.4.1 and Section 2.4.4.2.

## Handling of missing data for categorical efficacy endpoints

See Section 2.4.4.2.

### 2.5.4 Windows for time points /Measurements for analyses

The following steps will decide how the scheduled and/or unscheduled visits will be used in the analyses for efficacy variables and the by-visit summaries for safety variables (clinical laboratory data in Section 2.1.4.4 and vital signs in Section 2.1.4.5).

Step 1 A scheduled measurement will be used if it is available; otherwise, an unscheduled measurement (including the end of treatment/study visit for those prematurely discontinued) will be used if it happens to be on the same date as the date of the scheduled visit.

Step 2 After Step 1, if there are still no measurement for a given parameter at a scheduled visit, the analysis window below (Table 4) will be applied to re-allocate a post-baseline unscheduled measurement to a scheduled measurement.

Table 4 - Analyses window definition

| Targeted study day | Analysis window in study days |
|--------------------|---------------------------------------------|
| 28 | 2 to 55 |
| 84 | 56 to 104 |
| 126 | 105 to 153 |
| 182 | 154 to 227 |
| 273 | 228 to 318 |
| 364 | 319 to 409 |
| 455 | 410 to 502 |
| 551 | ≥503 |
| | 28<br>84<br>126<br>182<br>273<br>364<br>455 |

Study days are calculated from the day of first administration of double-blind IMP; the day of first administration of IMP (or the day of randomization if not exposed) is Day 1.

After applying the above time windows, if multiple assessments are associated to the same time point, the closest from the targeted study day will be used. In case of equality, the last measurement will be used. Re-allocated scheduled visits (ie, visit numbers) should be sequential if ordered by the date of measurement.

After Step 2, if there are still no measurement for a given parameter at a scheduled visit, data is considered missing for efficacy analyses, where multiple imputation would be applied as appropriately as described in Section 2.4.4.

## Reference day

The reference day for the calculation of extent of exposure, time to onset, and relative days will be the day of the first administration of double-blind IMP or the day of randomization if not exposed to double-blind IMP, denoted as Day 1.

## Baseline definition for efficacy/safety data

For the safety analyses, the baseline for a given parameter is defined as the last available measurement (or the average of all measurements for creatinine and eGFR), including unscheduled assessments, assessed prior to the first administration of double-blind IMP. For the efficacy analyses, the baseline for a given parameter is defined as the last available measurement (or the average of all measurements for creatinine and eGFR), including unscheduled assessments, assessed prior to the first administration of double-blind IMP or the last available value (or the average of all measurements for creatinine and eGFR) before randomization if not treated with double-blind IMP.

## Summary statistics by visit for continuous efficacy endpoints

Summary statistics (number, mean, SD, SE, minimum, median, maximum) of continuous efficacy endpoints (observed data and change from baseline) will be provided at scheduled visits as per protocol. Summaries showing data by visit will be presented according to the visit number (or re-allocated visit number) and labeled with the targeted approximate day/week.

#### Last on-treatment value for laboratory variables and vital signs

The last on-treatment value is the final measurement assessed during the treatment epoch, regardless of the introduction of rescue therapy, including measurements at unscheduled visits. Please see details in Section 2.1.4 and Section 2.4.5.

#### Display of safety data by visit (laboratory variables and vital signs)

Descriptive statistics (number, mean, SD, minimum, median, maximum) of quantitative laboratory variables and vital signs (observed data and change from baseline) during the TEAE period will be provided at scheduled visits. In addition, these summaries will also include a row for the 'last value on-treatment' to describe the last available on-treatment value (see above). Summaries showing data by visit will be presented according to the visit number (or re-allocated visit number, see Section 2.5.4) and labeled with the targeted approximate day/week.

As specified in the study protocol, laboratory data from scheduled visits are reported by central laboratories. The local results will not be used in the efficacy analyses or in the definition of baseline for both safety and efficacy analyses. In the safety analyses, for parameters with PCSA defined based on normal range, local results will only be used in the PCSA summary if they are accompanied by a local laboratory normal range. For parameters with PCSA not defined based on normal range, local results will be used in the PCSA summary as appropriately.

When a patient has more than 1 measurement from the central laboratory for the same laboratory parameter on the same date, the average of the measurements will be used. For the same laboratory parameter, if a patient has more than 1 measurement on different dates for the same scheduled visit, the value closest to the date of the visit will be used for the scheduled visit. When the values for the same scheduled visit are equidistant, the last value should be used for the scheduled visit. Similar rules will be applicable to a patient who has more than 1 set of measurements for the same vital sign parameter (ie, SBP, DBP, or HR) on the same date.

## 26-week double blind core treatment period

The 26-week double-blind core treatment period is the time from first administration of double-blind IMP to the last administration of double-blind IMP on or before Visit 9/Week 26 (or Day 182 if Visit 9/Week 26 date is missing). This is for analyzing selected efficacy parameters (eg, rescued patients) during core treatment period.

## TEAE period for the 26-week double blind core treatment period

The TEAE period for core treatment period is (1) the time from the first administration of the double-blind IMP up to 10 days (1 day for hypoglycemia) after the last administration of IMP if the patient discontinued treatment on or before Visit 9 (or Day 182 if Visit 9 date is missing), or (2) the time from the first administration of the double-blind IMP to the administration at Visit 9/Week 26 (or Day 182 if Visit 9/Week 26 date is missing) if the patient remained treated beyond Visit 9/Week 26. This is for the purpose of safety analyses during the core treatment period.

#### Time to event analysis

For time to event analysis/KM plot, time to event (eg, treatment discontinuation, rescue therapy, hypoglycemia, etc) is defined as the number of days from the date of the first administration of double-blind IMP (or the date of randomization if not exposed) to the start date of the first occurrence of the event during the 79-week double-blind treatment period.

Patients who did not experience any event during the 79-week double-blind treatment period are considered censored observations. For time to treatment discontinuation/rescue therapy, censoring date is the date of EOT. For time to severe or documented hypoglycemia, censoring date is date of EOT+1 or date of EOS, whichever is the earliest. Date of EOS will be used if date of EOT is not available. Last contact date will be used if date of EOS is not available.

#### 2.5.5 Unscheduled visits

Unscheduled visit measurements of laboratory data, vital signs, and ECG will be used for computation of baseline, the last on-treatment value, PCSAs and the shift summaries for safety or efficacy. They will be included in the by-visit summaries if they are re-allocated to scheduled visits (see Section 2.5.4).

## 2.5.6 Pooling of centers for statistical analyses

Center will not be included in the statistical models for efficacy analyses. However, all centers within a country will be pooled, and country will be included as a fixed effect in a parametric statistical model (eg, ANCOVA etc) for primary and secondary efficacy endpoints. Countries with fewer than 5 randomized patients will be grouped, if patients from grouped countries are still fewer than 5, they will then be further grouped with the country with the country with the lowest number of patients that is 5 or more.

#### 2.5.7 Statistical technical issues

None.

# 3 INTERIM ANALYSIS

No formal interim analysis for efficacy is planned for this study. The study will not be terminated early for excellent efficacy.

An independent Data Monitoring Committee (DMC) will be used to monitor and assess the safety of patients from this trial through periodic review of the accumulated safety data provided by an independent statistical group. Related details are provided in separate documents (DMC charter and DMC SAP).

# 4 DATABASE LOCK

The database is planned to be locked approximately 4 weeks after the last patient last visit.

# 5 SOFTWARE DOCUMENTATION

All summaries and statistical analyses will be generated using SAS® version 9.2 or higher.

| 6 | R | F | F | F | R | F | N | C | E | S |
|---|---|---|---|---|---|---|---|---|---|---|
| • | | _ | | _ | | _ | | • | | v |

None.

COVANCE INC. CONFIDENTIAL

# 7 LIST OF APPENDICES

Appendix A Potentially clinically significant abnormalities criteria

Appendix B List of PTs for select EOSIs (MedDRA v22.0)

Appendix C Summary of statistical analyses

Appendix D Study flow chart

# Appendix A Potentially clinically significant abnormalities criteria

# CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES for phase 2/3 studies (oncology excepted) (From BTD-009536 May 21, 2014)

| Parameter | PCSA | Comments |
|---|---|---|
| Clinical Chemistry | | |
| ALT | By distribution analysis : >3 ULN | Enzymes activities must be expressed in ULN, not in IU/L. |
| | >5 ULN<br>>10 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | >20 ULN | Internal DILI WG Oct 2008. |
| | 720 OLIV | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| AST | By distribution analysis : >3 ULN | Enzymes activities must be expressed in ULN, not in IU/L. |
| | >5 ULN<br>>10 ULN | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | >20 ULN | Internal DILI WG Oct 2008. |
| | 25 52.1 | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| Alkaline Phosphatase | >1.5 ULN | Enzymes activities must be expressed in ULN, not in IU/L. |
| | | Concept paper on DILI – FDA draft Guidance Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| Total Bilirubin | >1.5 ULN<br>>2 ULN | Must be expressed in ULN, not in µmol/L or mg/L. Categories are cumulative. |
| | 72 OLIN | Concept paper on DILI – FDA draft Guidance<br>Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| Conjugated Bilirubin | >35% Total Bilirubin and TBILI>1.5 ULN | Conjugated bilirubin dosed on a case-by-case basis. |
| ALT and Total Bilirubin | ALT>3 ULN and TBILI>2 ULN | Concept paper on DILI – FDA draft Guidance<br>Oct 2007. |
| | | Internal DILI WG Oct 2008. |
| | | To be counted within a same treatment<br>phase, whatever the interval between<br>measurement. |
| CPK | >3 ULN | FDA Feb 2005. |

## CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

| Parameter | PCSA | Comments |
|---|---|---|
| | >10 ULN | Am J Cardiol April 2006. |
| | | Categories are cumulative. |
| | | First row is mandatory. Rows following one mentioning zero can be deleted. |
| CLcr (mL/min) (Estimated creatinine clearance based on the Cokcroft-Gault equation) | <15 (end stage renal disease) ≥15 - <30 (severe decrease in GFR) ≥30 - < 60 (moderate decrease in GFR) ≥60 - <90 (mild decrease in GFR) ≥ 90 (normal GFR) | FDA draft Guidance 2010 Pharmacokinetics in patients with impaired renal function-study design, data analysis, and impact on dosing and labeling |
| eGFR (mL/min/1.73m2) | <15 (end stage renal disease) | FDA draft Guidance 2010 |
| (Estimate of GFR based on an MDRD equation) | ≥15 - <30 (severe decrease in GFR)<br>≥30 - < 60 (moderate decrease in GFR)<br>≥60 - <90 (mild decrease in GFR)<br>≥ 90 (normal GFR) | Pharmacokinetics in patients with impaired renal function-study design, data analysis, and impact on dosing and labeling |
| Creatinine | ≥150 µmol/L (Adults)<br>≥30% change from baseline<br>≥100% change from baseline | Benichou C., 1994. |
| Uric Acid | | Harrison- Principles of internal Medicine 17th |
| Hyperuricemia | >408 µmol/L | Ed., 2008. |
| Hypouricemia | <120 µmol/L | |
| Blood Urea Nitrogen | ≥17 mmol/L | |
| Chloride | <80 mmol/L | |
| | >115 mmol/L | |
| Sodium | ≤129 mmol/L<br>≥160 mmol/L | |
| Potassium | <3 mmol/L<br>≥5.5 mmol/L | FDA Feb 2005. |
| Total Cholesterol | ≥7.74 mmol/L | Threshold for therapeutic intervention. |
| Triglycerides | ≥4.6 mmol/L | Threshold for therapeutic intervention. |
| Lipasemia | ≥3 ULN | |
| Amylasemia | ≥3 ULN | |
| Glucose | | |
| Hypoglycaemia | ≤3.9 mmol/L and <lln< td=""><td>ADA May 2005.</td></lln<> | ADA May 2005. |
| Hyperglycaemia | ≥11.1 mmol/L (unfasted); ≥7 mmol/L (fasted) | ADA Jan 2008. |

## CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

| Parameter | PCSA | Comments |
|---|---|---|
| HbA1c | >8% | |
| Albumin | ≤25 g/L | |
| CRP | >2 ULN or >10 mg/L (if ULN not provided) | FDA Sept 2005. |
| Hematology | | |
| WBC | <3.0 Giga/L (Non-Black); <2.0 Giga/L (Black)<br>≥16.0 Giga/L | Increase in WBC: not relevant. To be interpreted only if no differential count available. |
| Lymphocytes | >4.0 Giga/L | |
| Neutrophils | <1.5 Giga/L (Non-Black);<1.0 Giga/L (Black) | International Consensus meeting on drug-<br>induced blood cytopenias, 1991.<br>FDA criteria. |
| Monocytes | >0.7 Giga/L | |
| Basophils | >0.1 Giga/L | |
| Eosinophils | >0.5 Giga/L or >ULN (if ULN≥0.5 Giga/L) | Harrison- Principles of internal Medicine 17th Ed., 2008. |
| Hemoglobin | ≤115 g/L (Male); ≤95 g/L (Female)<br>≥185 g/L (Male); ≥165 g/L (Female)<br>Decrease from Baseline ≥20 g/L | Criteria based upon decrease from baseline are more relevant than based on absolute value. Other categories for decrease from baseline can be used (≥30 g/L, ≥40 g/L, ≥50 g/L). |
| Hematocrit | ≤0.37 v/v (Male) ; ≤0.32 v/v (Female)<br>≥0.55 v/v (Male) ; ≥0.5 v/v (Female) | _50 g/L). |
| RBC | ≥6 Tera/L | Unless specifically required for particular drug development, the analysis is redundant with that of Hb. Otherwise, consider FDA criteria. |
| Platelets | <100 Giga/L<br>≥700 Giga/L | International Consensus meeting on drug-<br>induced blood cytopenias, 1991. |
| Urinalysis | | |
| pH | ≤4.6<br>≥8 | |
| Vital signs | | |
| HR | ≤50 bpm and decrease from baseline ≥20 bpm | To be applied for all positions (including missing) except STANDING. |

## CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

| Parameter | PCSA | Comments |
|---|---|---|
| | ≥120 bpm and increase from baseline≥20 bpm | |
| SBP | ≤95 mmHg and decrease from baseline ≥20mmHg<br>≥160 mmHg and increase from baseline ≥20 mmHg | To be applied for all positions (including missing) except STANDING. |
| DBP | ≤45 mmHg and decrease from baseline ≥10 mmHg<br>≥110 mmHg and increase from baseline ≥10 mmHg | To be applied for all positions (including missing) except STANDING. |
| Orthostatic Hypotension<br>Orthostatic SDB<br>Orthostatic DBP | ≤-20 mmHg<br>≤-10 mmHg | |
| Weight | ≥5% increase from baseline<br>≥5% decrease from baseline | FDA Feb 2007. |
| ECG | | Ref.: ICH E14 guidance (2005) and E14 Q&A (2012), and Cardiac Safety Research Consortium White Paper on PR and QRS (Nada et al. Am Heart J. 2013; 165(4): 489-500) |
| HR | <50 bpm<br><50 bpm and decrease from baseline ≥20 bpm<br><40 bpm<br><40 bpm and decrease from baseline ≥20 bpm<br><30 bpm<br><30 bpm and decrease from baseline ≥20 bpm | Categories are cumulative |
| | >90 bpm >90 bpm and increase from baseline ≥20bpm >100 bpm >100 bpm and increase from baseline ≥20bpm >120 bpm >120 bpm and increase from baseline ≥20 bpm | Categories are cumulative |
| PR | >200 ms >200 ms and increase from baseline ≥25% > 220 ms >220 ms and increase from baseline ≥25% > 240 ms > 240 ms and increase from baseline ≥25% | Categories are cumulative |
| QRS | >110 ms | Categories are cumulative |

## CRITERIA for POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITIES

| Parameter | PCSA | Comments |
|---|---|---|
| | >110 msec and increase from baseline ≥25% | |
| | >120 ms | |
| | >120 ms and increase from baseline ≥25% | |
| QT | >500 ms | |
| QTc | Absolute values (ms) | To be applied to any kind of QT correction formula. |
| | >450 ms | Absolute values categories are cumulative |
| | >480 ms | |
| | >500 ms | QTc >480 ms and \( \Delta\text{Tc} >60 \) ms are the 2 PCSA categories to be identified in individual |
| | Increase from baseline | subjects/patients listings. |
| | Increase from baseline ]30-60] ms | |
| | Increase from baseline >60 ms | |

# Appendix B List of PTs for select EOSIs (MedDRA v22.0)

| Genital Mycotic Infections 10014074 Balanitis candida Genital Mycotic Infections 10018143 Genital candidiasis Genital Mycotic Infections 10047784 Vulvovaginal candidiasis Genital Mycotic Infections 10064899 Vulvovaginal infection fungal Genital Mycotic Infections 10064899 Vulvovaginal mycotic infection Genital Mycotic Infections 10065582 Urogenital infection fungal Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 100717209 Candida cervicitis Urinary tract infections 10011791 Cystitis escherichia Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10037534 Pyelitis Urinary tract infections 10037594 Pyelitis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10038351 Renal abscess Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046424 Urethritis chlamydial Urinary tract infections 10046480 Urethritis chlamydial Urinary tract infections 10046480 Urethritis chlamydial Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046870 Urosepsis Urinary tract infections 10046870 Urosepsis Urinary tract infections 1004880 Urosepsis Urinary tract infections 1004890 Uros | EOSI | Preferred<br>Term Code | Preferred Term |
|---|---|---|---|
| Genital Mycotic Infections 10047784 Vulvovaginal candidiasis Genital Mycotic Infections 10064899 Vulvovaginal mycotic infection Genital Mycotic Infections 10064899 Vulvovaginal mycotic infection Genital Mycotic Infections 10065822 Urogenital infection fungal Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10071209 Candida cervicitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011790 Cystitis klebsiella Urinary tract infections 10011799 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelltis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis acute Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10034828 Tuberculosis of genitourinary system Urinary tract infections 1004828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046482 Urethritis Urinary tract infections 10046480 Urethritis Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046890 Urethritis ureaplasmal | Genital Mycotic Infections | 10004074 | Balanitis candida |
| Genital Mycotic Infections 10061180 Genital infection fungal Genital Mycotic Infections 10064899 Vulvovaginal mycotic infection Genital Mycotic Infections 10065582 Urogenital infection fungal Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10079521 Fungal balanitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011790 Cystitis secherichia Urinary tract infections 10011791 Cystitis secherichia Urinary tract infections 10011792 Cystitis selbasiella Urinary tract infections 10011793 Cystitis selbasiella Urinary tract infections 10011795 Fungal cystitis Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10037544 Kidney infection Urinary tract infections 10037594 Pyellitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037633 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 10046480 Urethritis Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046870 Urinary tract infection Urinary tract infections 10046870 Urinary tract infection Urinary tract infections 10046870 Urinary tract infections 1004690 Urinary tract infections 1004690 Urinary tract infection | Genital Mycotic Infections | 10018143 | Genital candidiasis |
| Genital Mycotic Infections 10064899 Vulvovaginal mycotic infection Genital Mycotic Infections 10065582 Urogenital infection fungal Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10079521 Fungal balanitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis secherichia Urinary tract infections 10011790 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10037542 Fungal cystitis Urinary tract infections 10037594 Pyellits Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections | Genital Mycotic Infections | 10047784 | Vulvovaginal candidiasis |
| Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10079521 Fungal balanitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 100117525 Fungal cystitis Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10037524 Kidney infection Urinary tract infections 10037524 Pyelitis Urinary tract infections 10037524 Pyelitis Urinary tract infections 10037526 Pyelonephritis Urinary tract infections 10037527 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10038351 Renal abscess Urinary tract infections 10048428 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis chlamydial Urinary tract infections 10046480 Urethritis infections Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 1004830 Tuberoundinary tract infections 1004680 Urethritis ureaplasmal Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 1004830 Tubulointerstitial nephritis Urinary tract infections 1004830 Urogenital trichomoniasis Urinary tract infections 1004830 Urogenital trichomoniasis Urinary tract infections 1004830 Urogenital trichomoniasis Urinary tract infections 1004830 Urinary tract infections 1004830 Urogenital trichomoniasis Urinary tract infections 1004830 Urinary tract inf | Genital Mycotic Infections | 10061180 | Genital infection fungal |
| Genital Mycotic Infections 10071209 Candida cervicitis Genital Mycotic Infections 10079521 Fungal balanitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis secherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 1003424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis cute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037633 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 10044828 Urethritis Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046480 Urethritis gonococcal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046571 Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10046870 Urosepsis Urinary tract infections 10048302 Cystitis glandularis Urinary tract infections 10049099 Urinary tract infection fungal Urinary tract infections 10049099 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Genital Mycotic Infections | 10064899 | Vulvovaginal mycotic infection |
| Genital Mycotic Infections 10079521 Fungal balanitis Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis secherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011797 Cystitis pseudomonal Urinary tract infections 10011795 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyenephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 1004828 Tuberculosis of genitourinary system Urinary tract infections 10044828 Urethral abscess Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046480 Urethritis gonococcal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 1004900 Pyelocystitis | Genital Mycotic Infections | 10065582 | Urogenital infection fungal |
| Urinary tract infections 10011781 Cystitis Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 1004482 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection enterococcal Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 1004883 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 1004900 Pyelocystitis | Genital Mycotic Infections | 10071209 | Candida cervicitis |
| Urinary tract infections 10011790 Cystitis escherichia Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 1004828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046481 Urethritis chlamydial Urinary tract infections 10046482 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046571 Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 1004900 Pyelocystitis | Genital Mycotic Infections | 10079521 | Fungal balanitis |
| Urinary tract infections 10011797 Cystitis klebsiella Urinary tract infections 10011799 Cystitis pseudomonal Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis chlamydial Urinary tract infections 10046482 Urethritis chlamydial Urinary tract infections 10046483 Urethritis chlamydial Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection 10046571 Urinary tract infection 10046571 Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048905 Urinary tract infection fungal Urinary tract infections 1004905 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10011781 | Cystitis |
| Urinary tract infections Urinary tract infecti | Urinary tract infections | 10011790 | Cystitis escherichia |
| Urinary tract infections 10017525 Fungal cystitis Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046482 Urethritis gonococcal Urinary tract infections 10046483 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046480 Urethritis ureaplasmal Urinary tract infections 10046671 Urinary tract infection Urinary tract infections 10046572 Urinary tract infection Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 1004837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10011797 | Cystitis klebsiella |
| Urinary tract infections 10018185 Genitourinary chlamydia infection Urinary tract infections 10023424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 1004828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046482 Urethritis chlamydial Urinary tract infections 10046483 Urethritis gonococcal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 1004837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10011799 | Cystitis pseudomonal |
| Urinary tract infections 1003424 Kidney infection Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037597 Pyelonephritis acute Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 1004828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046482 Urethritis chlamydial Urinary tract infections 10046483 Urethritis gonococcal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10017525 | Fungal cystitis |
| Urinary tract infections 10037584 Pyelitis Urinary tract infections 10037596 Pyelonephritis Urinary tract infections 10037601 Pyelonephritis chronic Urinary tract infections 10037603 Pyelonephritis mycoplasmal Urinary tract infections 10037653 Pyonephrosis Urinary tract infections 10038351 Renal abscess Urinary tract infections 10044828 Tuberculosis of genitourinary system Urinary tract infections 10046424 Urethral abscess Urinary tract infections 10046480 Urethritis Urinary tract infections 10046482 Urethritis chlamydial Urinary tract infections 10046483 Urethritis ureaplasmal Urinary tract infections 10046490 Urethritis ureaplasmal Urinary tract infections 10046571 Urinary tract infection Urinary tract infections 10046572 Urinary tract infection enterococcal Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary t | Urinary tract infections | 10018185 | Genitourinary chlamydia infection |
| Urinary tract infections10037596PyelonephritisUrinary tract infections10037597Pyelonephritis acuteUrinary tract infections10037601Pyelonephritis chronicUrinary tract infections10037603Pyelonephritis mycoplasmalUrinary tract infections10037653PyonephrosisUrinary tract infections10038351Renal abscessUrinary tract infections1004828Tuberculosis of genitourinary systemUrinary tract infections10044828Urethral abscessUrinary tract infections10046424UrethritisUrinary tract infections10046480Urethritis chlamydialUrinary tract infections10046482Urethritis gonococcalUrinary tract infections10046483Urethritis ureaplasmalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10023424 | Kidney infection |
| Urinary tract infections10037597Pyelonephritis acuteUrinary tract infections10037601Pyelonephritis chronicUrinary tract infections10037603Pyelonephritis mycoplasmalUrinary tract infections10037653PyonephrosisUrinary tract infections10038351Renal abscessUrinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037584 | Pyelitis |
| Urinary tract infections10037601Pyelonephritis chronicUrinary tract infections10037603Pyelonephritis mycoplasmalUrinary tract infections10037653PyonephrosisUrinary tract infections10038351Renal abscessUrinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037596 | Pyelonephritis |
| Urinary tract infections10037603Pyelonephritis mycoplasmalUrinary tract infections10037653PyonephrosisUrinary tract infections10038351Renal abscessUrinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037597 | Pyelonephritis acute |
| Urinary tract infections10037653PyonephrosisUrinary tract infections10038351Renal abscessUrinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037601 | Pyelonephritis chronic |
| Urinary tract infections10038351Renal abscessUrinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037603 | Pyelonephritis mycoplasmal |
| Urinary tract infections10044828Tuberculosis of genitourinary systemUrinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10037653 | Pyonephrosis |
| Urinary tract infections10046424Urethral abscessUrinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10038351 | Renal abscess |
| Urinary tract infections10046480UrethritisUrinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10044828 | Tuberculosis of genitourinary system |
| Urinary tract infections10046482Urethritis chlamydialUrinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10046424 | Urethral abscess |
| Urinary tract infections10046483Urethritis gonococcalUrinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10046480 | Urethritis |
| Urinary tract infections10046490Urethritis ureaplasmalUrinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10046482 | Urethritis chlamydial |
| Urinary tract infections10046571Urinary tract infectionUrinary tract infections10046572Urinary tract infection enterococcalUrinary tract infections10046704Urogenital trichomoniasisUrinary tract infections10048302Tubulointerstitial nephritisUrinary tract infections10048709UrosepsisUrinary tract infections10048837Cystitis glandularisUrinary tract infections10049059Urinary tract infection fungalUrinary tract infections10049100Pyelocystitis | Urinary tract infections | 10046483 | Urethritis gonococcal |
| Urinary tract infections 10046572 Urinary tract infection enterococcal Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10046490 | Urethritis ureaplasmal |
| Urinary tract infections 10046704 Urogenital trichomoniasis Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10046571 | Urinary tract infection |
| Urinary tract infections 10048302 Tubulointerstitial nephritis Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10046572 | Urinary tract infection enterococcal |
| Urinary tract infections 10048709 Urosepsis Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10046704 | Urogenital trichomoniasis |
| Urinary tract infections 10048837 Cystitis glandularis Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10048302 | Tubulointerstitial nephritis |
| Urinary tract infections 10049059 Urinary tract infection fungal Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10048709 | Urosepsis |
| Urinary tract infections 10049100 Pyelocystitis | Urinary tract infections | 10048837 | Cystitis glandularis |
| | Urinary tract infections | 10049059 | Urinary tract infection fungal |
| Urinary tract infections 10051250 Ureteritis | Urinary tract infections | 10049100 | Pyelocystitis |
| | Urinary tract infections | 10051250 | Ureteritis |

| Urinary tract infections | 10051350 | Cytomegalovirus urinary tract infection |
|---|---|---|
| Urinary tract infections | 10051959 | Urinary bladder abscess |
| Urinary tract infections | 10052238 | Escherichia urinary tract infection |
| Urinary tract infections | 10054088 | Urinary tract infection bacterial |
| Urinary tract infections | 10056351 | Emphysematous cystitis |
| Urinary tract infections | 10058523 | Bladder candidiasis |
| Urinary tract infections | 10058596 | Renal cyst infection |
| Urinary tract infections | 10059517 | Bacterial pyelonephritis |
| Urinary tract infections | 10061181 | Genitourinary tract gonococcal infection |
| Urinary tract infections | 10061182 | Genitourinary tract infection |
| Urinary tract infections | 10061395 | Ureter abscess |
| Urinary tract infections | 10062279 | Urinary tract infection pseudomonal |
| Urinary tract infections | 10062280 | Urinary tract infection staphylococcal |
| Urinary tract infections | 10064825 | Urinary tract infection viral |
| Urinary tract infections | 10064921 | Urinary tract inflammation |
| Urinary tract infections | 10065197 | Cystitis viral |
| Urinary tract infections | 10065198 | Cystitis bacterial |
| Urinary tract infections | 10065199 | Cystitis helminthic |
| Urinary tract infections | 10065213 | Pyelonephritis viral |
| Urinary tract infections | 10065214 | Pyelonephritis fungal |
| Urinary tract infections | 10065582 | Urogenital infection fungal |
| Urinary tract infections | 10065583 | Urogenital infection bacterial |
| Urinary tract infections | 10066757 | Urinary tract abscess |
| Urinary tract infections | 10068822 | Emphysematous pyelonephritis |
| Urinary tract infections | 10070300 | Streptococcal urinary tract infection |
| Urinary tract infections | 10074409 | Escherichia pyelonephritis |
| Urinary tract infections | 10075063 | Urethritis mycoplasmal |
| Urinary tract infections | 10078665 | Bacterial urethritis |
| Urinary tract infections | 10081163 | Fungal urethritis |
| Urinary tract infections | 10081262 | Candida urethritis |
| Urinary tract infections | 10082040 | Nephritis bacterial |
| Volume depletion | 10005697 | Blood osmolarity increased |
| Volume depletion | 10005731 | Blood pressure ambulatory decreased |
| Volume depletion | 10005734 | Blood pressure decreased |
| Volume depletion | 10005737 | Blood pressure diastolic decreased |
| Volume depletion | 10005748 | Blood pressure immeasurable |
| Volume depletion | 10005758 | Blood pressure systolic decreased |
| Volume depletion | 10005761 | Blood pressure systolic inspiratory decreased |
| Volume depletion | 10007979 | Central venous pressure decreased |
| Volume depletion | 10009192 | Circulatory collapse |
| Volume depletion | 10012174 | Dehydration |
| Volume depletion | 10013578 | Dizziness postural |

| Volume depletion | 10021097 | Hypotension |
|---|---|---|
| Volume depletion | 10021137 | Hypovolaemia |
| Volume depletion | 10021138 | Hypovolaemic shock |
| Volume depletion | 10026983 | Mean arterial pressure decreased |
| Volume depletion | 10031127 | Orthostatic hypotension |
| Volume depletion | 10036653 | Presyncope |
| Volume depletion | 10037327 | Pulmonary arterial wedge pressure decreased |
| Volume depletion | 10042772 | Syncope |
| Volume depletion | 10046640 | Urine flow decreased |
| Volume depletion | 10047235 | Venous pressure decreased |
| Volume depletion | 10047239 | Venous pressure jugular decreased |
| Volume depletion | 10047689 | Volume blood decreased |
| Volume depletion | 10050760 | Blood urea nitrogen/creatinine ratio increased |
| Volume depletion | 10050905 | Decreased ventricular preload |
| Volume depletion | 10053356 | Blood pressure orthostatic decreased |
| Volume depletion | 10059895 | Urine output decreased |
| Volume depletion | 10060089 | Left ventricular end-diastolic pressure decreased |
| Volume depletion | 10060231 | Pulmonary arterial pressure decreased |
| Volume depletion | 10063080 | Postural orthostatic tachycardia syndrome |
| Volume depletion | 10063927 | Orthostatic intolerance |
| Volume depletion | 10066077 | Diastolic hypotension |
| Volume depletion | 10069431 | Orthostatic heart rate response increased |
| Volume depletion | 10069583 | Pulse volume decreased |
| Volume depletion | 10072370 | Prerenal failure |
| Pancreatitis | 10033625 | Pancreatic haemorrhage |
| Pancreatitis | 10033635 | Pancreatic pseudocyst |
| Pancreatitis | 10033636 | Pancreatic pseudocyst drainage |
| Pancreatitis | 10033645 | Pancreatitis |
| Pancreatitis | 10033647 | Pancreatitis acute |
| Pancreatitis | 10033649 | Pancreatitis chronic |
| Pancreatitis | 10033650 | Pancreatitis haemorrhagic |
| Pancreatitis | 10033654 | Pancreatitis necrotising |
| Pancreatitis | 10033657 | Pancreatitis relapsing |
| Pancreatitis | 10048984 | Pancreatic abscess |
| Pancreatitis | 10052400 | Oedematous pancreatitis |
| Pancreatitis | 10056277 | Pancreatorenal syndrome |
| Pancreatitis | 10056975 | Pancreatic phlegmon |
| Pancreatitis | 10056976 | Hereditary pancreatitis |
| Pancreatitis | 10056977 | Alcoholic pancreatitis |
| Pancreatitis | 10058096 | Pancreatic necrosis |
| Pancreatitis | 10065189 | Pancreatitis helminthic |
| Pancreatitis | 10066127 | Ischaemic pancreatitis |

Date of Issue: 19 February 2020

Covance Study ID:000000154257

| Venous thrombotic events | 10066881 | Deep vein thrombosis postoperative |
|---|---|---|
| Venous thrombotic events | 10067270 | Thrombosis corpora cavernosa |
| Venous thrombotic events | 10069909 | Metastatic pulmonary embolism |
| Venous thrombotic events | 10072059 | Ovarian vein thrombosis |
| Venous thrombotic events | 10074349 | Ophthalmic vein thrombosis |
| Venous thrombotic events | 10077623 | Portosplenomesenteric venous thrombosis |
| Venous thrombotic events | 10077829 | Visceral venous thrombosis |
| Venous thrombotic events | 10078810 | Hepatic vein embolism |
| Thyroid cancer | 10002240 | Anaplastic thyroid cancer |
| Thyroid cancer | 10016935 | Follicular thyroid cancer |
| Thyroid cancer | 10027105 | Medullary thyroid cancer |
| Thyroid cancer | 10033701 | Papillary thyroid cancer |
| Thyroid cancer | 10043744 | Thyroid neoplasm |
| Thyroid cancer | 10055107 | Thyroid cancer metastatic |
| Thyroid cancer | 10066136 | Huerthle cell carcinoma |
| Thyroid cancer | 10066474 | Thyroid cancer |
| Thyroid cancer | 10070567 | Thyroid cancer stage 0 |
| Thyroid cancer | 10071027 | Thyroid cancer stage I |
| Thyroid cancer | 10071028 | Thyroid cancer stage II |
| Thyroid cancer | 10071029 | Thyroid cancer stage III |
| Thyroid cancer | 10071030 | Thyroid cancer stage IV |
| Thyroid cancer | 10072162 | Thyroid cancer recurrent |
| Thyroid cancer | 10072613 | Thyroid B-cell lymphoma |
| Thyroid cancer | 10073153 | Familial medullary thyroid cancer |
| Thyroid cancer | 10076603 | Poorly differentiated thyroid carcinoma |
| Renal cell cancer | 10038389 | Renal cancer |
| Renal cell cancer | 10038390 | Renal cancer recurrent |
| Renal cell cancer | 10038391 | Renal cancer stage I |
| Renal cell cancer | 10038392 | Renal cancer stage II |
| Renal cell cancer | 10038393 | Renal cancer stage III |
| Renal cell cancer | 10038394 | Renal cancer stage IV |
| Renal cell cancer | 10038410 | Renal cell carcinoma recurrent |
| Renal cell cancer | 10038411 | Renal cell carcinoma stage I |
| Renal cell cancer | 10038412 | Renal cell carcinoma stage II |
| Renal cell cancer | 10038413 | Renal cell carcinoma stage III |
| Renal cell cancer | 10038414 | Renal cell carcinoma stage IV |
| Renal cell cancer | 10050018 | Renal cancer metastatic |
| Renal cell cancer | 10050513 | Metastatic renal cell carcinoma |
| Renal cell cancer | 10061482 | Renal neoplasm |
| Renal cell cancer | 10067944 | Hereditary leiomyomatosis renal cell carcinoma |
| Renal cell cancer | 10067946 | Renal cell carcinoma |
| Renal cell cancer | 10073251 | Clear cell renal cell carcinoma |

| Renal cell cancer | 10078493 | Papillary renal cell carcinoma |
|---|---|---|
| Pancreatic cancer | 10018404 | Glucagonoma |
| Pancreatic cancer | 10022498 | Insulinoma |
| Pancreatic cancer | 10025997 | Malignant neoplasm of islets of Langerhans |
| Pancreatic cancer | 10029341 | Neurotensinoma |
| Pancreatic cancer | 10033609 | Pancreatic carcinoma |
| Pancreatic cancer | 10033610 | Pancreatic carcinoma metastatic |
| Pancreatic cancer | 10033613 | Pancreatic carcinoma recurrent |
| Pancreatic cancer | 10041329 | Somatostatinoma |
| Pancreatic cancer | 10047430 | Vipoma |
| Pancreatic cancer | 10051709 | Gastrinoma malignant |
| Pancreatic cancer | 10052747 | Adenocarcinoma pancreas |
| Pancreatic cancer | 10055006 | Pancreatic sarcoma |
| Pancreatic cancer | 10055007 | Carcinoid tumour of the pancreas |
| Pancreatic cancer | 10059320 | Pancreatic carcinoma stage 0 |
| Pancreatic cancer | 10059321 | Pancreatic carcinoma stage I |
| Pancreatic cancer | 10059322 | Pancreatic carcinoma stage II |
| Pancreatic cancer | 10059323 | Pancreatic carcinoma stage III |
| Pancreatic cancer | 10059326 | Pancreatic carcinoma stage IV |
| Pancreatic cancer | 10061902 | Pancreatic neoplasm |
| Pancreatic cancer | 10067517 | Pancreatic neuroendocrine tumour |
| Pancreatic cancer | 10068909 | Pancreatic neuroendocrine tumour metastatic |
| Pancreatic cancer | 10069345 | Solid pseudopapillary tumour of the pancreas |
| Pancreatic cancer | 10073363 | Acinar cell carcinoma of pancreas |
| Pancreatic cancer | 10073364 | Ductal adenocarcinoma of pancreas |
| Pancreatic cancer | 10073365 | Intraductal papillary-mucinous carcinoma of pancreas |
| Pancreatic cancer | 10073367 | Pancreatoblastoma |
| Bladder cancer | 10004986 | Bladder adenocarcinoma recurrent |
| Bladder cancer | 10004987 | Bladder adenocarcinoma stage 0 |
| Bladder cancer | 10004988 | Bladder adenocarcinoma stage I |
| Bladder cancer | 10004989 | Bladder adenocarcinoma stage II |
| Bladder cancer | 10004990 | Bladder adenocarcinoma stage III |
| Bladder cancer | 10004991 | Bladder adenocarcinoma stage IV |
| Bladder cancer | 10004992 | Bladder adenocarcinoma stage unspecified |
| Bladder cancer | 10005003 | Bladder cancer |
| Bladder cancer | 10005005 | Bladder cancer recurrent |
| Bladder cancer | 10005006 | Bladder cancer stage 0, with cancer in situ |
| Bladder cancer | 10005007 | Bladder cancer stage 0, without cancer in situ |
| Bladder cancer | 10005008 | Bladder cancer stage I, with cancer in situ |
| Bladder cancer | 10005009 | Bladder cancer stage I, without cancer in situ |
| Bladder cancer | 10005010 | Bladder cancer stage II |

| Bladder cancer | 10005011 | Bladder cancer stage III |
|---|---|---|
| Bladder cancer | 10005012 | Bladder cancer stage IV |
| Bladder cancer | 10005056 | Bladder neoplasm |
| Bladder cancer | 10005075 | Bladder squamous cell carcinoma recurrent |
| Bladder cancer | 10005076 | Bladder squamous cell carcinoma stage 0 |
| Bladder cancer | 10005077 | Bladder squamous cell carcinoma stage I |
| Bladder cancer | 10005078 | Bladder squamous cell carcinoma stage II |
| Bladder cancer | 10005079 | Bladder squamous cell carcinoma stage III |
| Bladder cancer | 10005080 | Bladder squamous cell carcinoma stage IV |
| Bladder cancer | 10005081 | Bladder squamous cell carcinoma stage |
| | | unspecified |
| Bladder cancer | 10005084 | Bladder transitional cell carcinoma |
| Bladder cancer | 10051690 | Urinary bladder sarcoma |
| Bladder cancer | 10057352 | Metastatic carcinoma of the bladder |
| Bladder cancer | 10066749 | Bladder transitional cell carcinoma stage 0 |
| Bladder cancer | 10066750 | Bladder transitional cell carcinoma recurrent |
| Bladder cancer | 10066751 | Bladder transitional cell carcinoma stage I |
| Bladder cancer | 10066752 | Bladder transitional cell carcinoma stage IV |
| Bladder cancer | 10066753 | Bladder transitional cell carcinoma stage II |
| Bladder cancer | 10066754 | Bladder transitional cell carcinoma stage III |
| Bladder cancer | 10071664 | Bladder transitional cell carcinoma metastatic |
| Bladder cancer | 10078341 | Neuroendocrine carcinoma of the bladder |
| Potentially leading to amputation | 10003084 | Areflexia |
| Potentially leading to amputation | 10003178 | Arterial thrombosis |
| Potentially leading to amputation | 10003210 | Arteriosclerosis |
| Potentially leading to amputation | 10003222 | Arteriosclerotic gangrene |
| Potentially leading to amputation | 10006784 | Burning sensation |
| Potentially leading to amputation | 10007904 | Cellulitis enterococcal |
| Potentially leading to amputation | 10007905 | Cellulitis gangrenous |
| Potentially leading to amputation | 10007921 | Cellulitis staphylococcal |
| Potentially leading to amputation | 10007922 | Cellulitis streptococcal |
| Potentially leading to amputation | 10012174 | Dehydration |
| Potentially leading to amputation | 10012665 | Diabetic gangrene |
| Potentially leading to amputation | 10012679 | Diabetic neuropathic ulcer |
| Potentially leading to amputation | 10012680 | Diabetic neuropathy |
| Potentially leading to amputation | 10017711 | Gangrene |
| Potentially leading to amputation | 10020937 | Hypoaesthesia |
| Potentially leading to amputation | 10021137 | Hypovolaemia |
| Potentially leading to amputation | 10021519 | Impaired healing |
| Potentially leading to amputation | 10021784 | Infected skin ulcer |
| Potentially leading to amputation | 10022562 | Intermittent claudication |
| Potentially leading to amputation | 10024774 | Localised infection |
| Potentially leading to amputation | 10028862 | Necrosis ischaemic |
| Potentially leading to amputation | 10029331 | Neuropathy peripheral |

| Potentially leading to amputation | 10031149 | Osteitis |
|---|---|---|
| Potentially leading to amputation | 10031252 | Osteomyelitis |
| Potentially leading to amputation | 10031253 | Osteomyelitis acute |
| Potentially leading to amputation | 10031256 | Osteomyelitis chronic |
| Potentially leading to amputation | 10031262 | Osteomyelitis salmonella |
| Potentially leading to amputation | 10031264 | Osteonecrosis |
| Potentially leading to amputation | 10033775 | Paraesthesia |
| Potentially leading to amputation | 10034568 | Peripheral coldness |
| Potentially leading to amputation | 10034576 | Peripheral ischaemia |
| Potentially leading to amputation | 10034620 | Peripheral sensory neuropathy |
| Potentially leading to amputation | 10034636 | Peripheral vascular disorder |
| Potentially leading to amputation | 10036155 | Poor peripheral circulation |
| Potentially leading to amputation | 10036410 | Postoperative wound infection |
| Potentially leading to amputation | 10040026 | Sensory disturbance |
| Potentially leading to amputation | 10040840 | Skin erosion |
| Potentially leading to amputation | 10040872 | Skin infection |
| Potentially leading to amputation | 10040943 | Skin ulcer |
| Potentially leading to amputation | 10042343 | Subcutaneous abscess |
| Potentially leading to amputation | 10043607 | Thrombosis |
| Potentially leading to amputation | 10048031 | Wound dehiscence |
| Potentially leading to amputation | 10048038 | Wound infection |
| Potentially leading to amputation | 10049927 | Dry gangrene |
| Potentially leading to amputation | 10050473 | Abscess limb |
| Potentially leading to amputation | 10050502 | Neuropathic ulcer |
| Potentially leading to amputation | 10051548 | Burn infection |
| Potentially leading to amputation | 10052428 | Wound |
| Potentially leading to amputation | 10052949 | Arterial therapeutic procedure |
| Potentially leading to amputation | 10053692 | Wound complication |
| Potentially leading to amputation | 10053716 | Wound necrosis |
| Potentially leading to amputation | 10054044 | Diabetic microangiopathy |
| Potentially leading to amputation | 10056340 | Diabetic ulcer |
| Potentially leading to amputation | 10056418 | Arterial bypass operation |
| Potentially leading to amputation | 10056673 | Peripheral sensorimotor neuropathy |
| Potentially leading to amputation | 10057518 | Peripheral artery angioplasty |
| Potentially leading to amputation | 10057525 | Peripheral artery occlusion |
| Potentially leading to amputation | 10058041 | Wound sepsis |
| Potentially leading to amputation | 10058042 | Wound abscess |
| Potentially leading to amputation | 10059245 | Angiopathy |
| Potentially leading to amputation | 10059385 | Extremity necrosis |
| Potentially leading to amputation | 10059442 | Wound infection staphylococcal |
| Potentially leading to amputation | 10059444 | Wound infection pseudomonas |
| Potentially leading to amputation | 10060734 | Diabetic foot |
| Potentially leading to amputation | 10060803 | Diabetic foot infection |
| Potentially leading to amputation | 10060963 | Arterial disorder |
| Potentially leading to amputation | 10060965 | Arterial stenosis |

| Potentially leading to amputation | 10061627 | Amputation |
|---|---|---|
| Potentially leading to amputation | 10061655 | Arterial graft |
| Potentially leading to amputation | 10061657 | Arterial stent insertion |
| Potentially leading to amputation | 10061666 | Autonomic neuropathy |
| Potentially leading to amputation | 10061815 | Diabetic vascular disorder |
| Potentially leading to amputation | 10062198 | Microangiopathy |
| Potentially leading to amputation | 10062255 | Soft tissue infection |
| Potentially leading to amputation | 10062585 | Peripheral arterial occlusive disease |
| Potentially leading to amputation | 10062599 | Arterial occlusive disease |
| Potentially leading to amputation | 10062610 | Ischaemic limb pain |
| Potentially leading to amputation | 10062932 | Wound treatment |
| Potentially leading to amputation | 10064250 | Staphylococcal osteomyelitis |
| Potentially leading to amputation | 10064601 | Iliac artery occlusion |
| Potentially leading to amputation | 10065237 | Osteomyelitis bacterial |
| Potentially leading to amputation | 10065239 | Osteomyelitis fungal |
| Potentially leading to amputation | 10065240 | Wound infection bacterial |
| Potentially leading to amputation | 10065242 | Wound infection fungal |
| Potentially leading to amputation | 10068653 | Bone abscess |
| Potentially leading to amputation | 10069379 | Peripheral arterial reocclusion |
| Potentially leading to amputation | 10072170 | Skin wound |
| Potentially leading to amputation | 10072557 | Peripheral artery restenosis |
| Potentially leading to amputation | 10072560 | Peripheral endarterectomy |
| Potentially leading to amputation | 10072561 | Peripheral artery bypass |
| Potentially leading to amputation | 10072562 | Peripheral artery stent insertion |
| Potentially leading to amputation | 10072563 | Peripheral artery stenosis |
| Potentially leading to amputation | 10072564 | Peripheral artery thrombosis |
| Potentially leading to amputation | 10074396 | Penetrating atherosclerotic ulcer |
| Potentially leading to amputation | 10075118 | Subperiosteal abscess |
| Potentially leading to amputation | 10075714 | Vasculitic ulcer |
| Potentially leading to amputation | 10076246 | Spontaneous amputation |

# Appendix C Summary of statistical analyses

## EFFICACY ANALYSIS

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other<br>analyses |
|---|---|---|---|---|---|
| Primary endpoint | | | | | |
| HbA1c: Change from<br>Baseline at Week 26 | ΙΠ | ANCOVA (with missing values imputed by the retrieved dropouts imputation method or by washout MI method under MNAR framework): treatment, randomization stratum (HbA1c /metformin use/ SBP at screening), and country as fixed effects, and baseline HbA1c value as a covariate | Tipping point analysis; | Subgroups: race,<br>ethnicity, age, gender,<br>baseline BMI,<br>baseline HbA1c,<br>baseline SBP,<br>metformin use at<br>screening, baseline<br>eGFR, Duration of<br>diabetes, and country | Summary statistics for observed values and changes from baseline by visit. Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit. By-visit summary and graph excluding measurements after rescue therapy. |
| Secondary endpoints | | | | | |
| FPG, body weight: Change from baseline to Week 26; SBP (for patients with Baseline SBP ≥130 mmHg, all patients): Change from Baseline to Week 12 | ITT | ANCOVA (with missing values imputed by the retrieved dropouts imputation method or by washout MI Method under MNAR framework): treatment, randomization stratum (HbA1c /metformin use / SBP at screening), and country as fixed effects, and baseline value as a covariate | No | No | Summary statistics for observed values and changes from baseline by visit. Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit. SBP will be summarized descriptively at each visit for those with baseline SBP ≥140 mmHg |
| Proportion of patients with<br>HbA1c <6.5%, <7.0% at<br>Week 26 | ІТТ | CMH method stratified on randomization strata (HbA1c /metformin use / SBP at | CMH method stratified on randomization strata (HbA1c /metformin use/ | No | By-visit summary and graphs of HbA <sub>1c</sub> responders (<6.5%, <7%). |
| FFCCR 20 | | screening), | SBP at screen: excluding | | By-visit frequency summary and graphs of HbA1c responders (<6.5%, <7%) |

| Endpoint | Analysis population | Primary<br>analysis | Supportive analysis | Subgroup<br>analysis | Other<br>analyses |
|---|---|---|---|---|---|
| | | | patients with baseline<br>HbA <sub>1c</sub> values <6.5% (for<br><6.5% responders) or<br><7% (for <7%<br>responders) respectively | | excluding patients with baseline $HbA_{1c}$ values <6.5% or <7% respectively. |
| Other endpoints | | | | | |
| SBP (for patients with<br>baseline SBP <130 mmHg),<br>DBP, Serum creatinine,<br>eGFR: change from Baseline | ΙΤΤ | Summary statistics for observed values and changes from baseline by visit. | No | No | Graphical presentations for mean changes from baseline (±SE) and mean values (±SE) by visit as appropriate. |
| Proportion of patients, with reduction in body weight by ≥2%, ≥5%, and ≥10% from Baseline; achieving SBP <130 mmHg with baseline SBP ≥130 mmHg; achieving DBP <80 mmHg with baseline DBP ≥80 mmHg | ΙΤΤ | By-visit frequency summary | No | No | By-visit graphical presentation as appropriate |
| Proportion of patients requiring rescue for hyperglycemia | | Summary statistics | No | No | KM plot; List of patients rescued |

# SAFETY ANALYSES

| Endpoint | Analysis Primary Supportive<br>Population analysis Analysis | | | Subgroup<br>analysis | Other analyses |
|---|---|---|---|---|---|
| Hypoglycemia | Safety | Follow safety guidelines Number (%) of patients with any hypoglycemia, severe hypoglycemia, documented symptomatic hypoglycemia during TEAE period, and incidence rates in 100 patient- years. | | Severe hypoglycemia or<br>documented symptomatic<br>hypoglycemia by subgroups:<br>race, age, gender, metformin use | KM plot time to first event of severe hypoglycemia or documented symptomatic hypoglycemia Documented symptomatic hypoglycemia maybe presented by <3.0 mmol/L (<54 mg/dL) as appropriate. |
| Adverse Events | Safety | Follow safety guidelines | No | Common TEAEs by subgroups: race, age, gender, baseline SBP, metformin use, baseline eGFR | To be updated for EOSI |
| Clinical laboratory data | Safety | Follow safety guidelines | Descriptive | No | No |
| Vital signs | Safety | Follow safety guidelines | Descriptive | No | No |
| ECG, Physical examination | Safety | Follow safety guidelines | Frequency summary | No | No |

# Appendix D Study flow chart

| | Screening | Period | Double-Blind Core Treatment Period <sup>a</sup> | | | | | | | | uble-B | Follow-up | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | | | | | | P | | | | | | | |
| VISIT | 1 | 2 | 3<br>Baseline | 4<br><b>2</b> | 5 | 6 <sup>€</sup> | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14<br><b>22</b> |
| Week | -4 | -2 | 0 | 1 | 4 | 8 | 12 | 18 | 26 | 39 | 52 | 65 | 79 | 81 |
| Day (window [days]) | | -14<br>(±3) | 1<br>(-) | 7<br>(±3) | 28<br>(±3) | 56<br>(±3) | 84<br>(±3) | 126<br>(±3) | 182<br>(±3) | 273<br>(±7) | 364<br>(±7) | 455<br>(±7) | 551<br>(-3 to +4) | 565<br>(±3) |
| Informed consent | Х | | | | | | | | | | | | | |
| Inclusion criteria | Х | | | | | | | | | | | | | |
| Exclusion criteria | х | Х | X | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | |
| Medical/Surgical History | Х | | | | | | | | | | | | | |
| Medication History | Х | | | | | | | | | | | | | |
| Body weight, height <sup>d</sup> | Х | Х | X | | Х | | Х | Х | Χ | Х | Х | Х | Х | |
| Vital signs <sup>e</sup> | Х | Х | Х | | X | | X | Х | Х | X | Х | Х | Х | |
| Physical Examination: | | | | | | | | | | | | | | |
| Complete | Х | | | | | | | | X | | | | Х | |
| Abbreviated <sup>f</sup> | | Х | X | | Х | | Х | Х | | Х | Х | Х | | |
| Diet & exercise instruction | | Х | Х | | | | | | Х | | Х | | Х | |
| Instruction on basic GU hygiene & hydration | | Х | Х | Х | Х | х | Х | X | х | Х | Х | Х | Х | |

| | Screening | Period | Dou | Double-Blind Core Treatment Perio | | | | eriod <sup>a</sup> | | Double-Blind Extension | | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Run-In | | | | | | | | | P | eriod <sup>b</sup> | | |
| VISIT | 1 | 2 | 3<br>Baseline | 4<br><b>2</b> | 5 | 6 <sup>€</sup> | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Week | -4 | -2 | 0 | 1 | 4 | 8 | 12 | 18 | 26 | 39 | 52 | 65 | 79 | 81 |
| Day (window [days]) | | -14<br>(±3) | 1<br>(-) | 7<br>(±3) | 28<br>(±3) | 56<br>(±3) | 84<br>(±3) | 126<br>(±3) | 182<br>(±3) | 273<br>(±7) | 364<br>(±7) | 455<br>(±7) | 551<br>(-3 to +4) | 565<br>(±3) |
| Interactive response technology (IRT) contact | Х | Х | Х | | X | | X | X | Х | Х | Х | Х | Х | Х |
| Randomization | | | Х | | | | | | | | | | | |
| Dispense glucose meter | | Х | | | | | | | | | | | | |
| Dispense diary | Х | Х | Х | | Х | | Х | Х | Х | Х | Х | Х | | |
| Collect/review diary | | Х | Х | | X | | X | X | X | X | X | Х | Х | |
| Instruction on diabetic ketoacidosis symptoms, glucose testing | | | х | х | Х | X | Х | X | х | Х | х | Х | Х | |
| Dispense IMP | | Х | Х | | Х | | Х | Х | Х | Х | Х | Х | | |
| IMP accounting & compliance | | | Х | | Х | | Х | Х | Х | Х | Х | Х | Х | |
| Concomitant Medication | Х | Х | Х | X | X | X | X | X | X | X | X | X | X | X |
| SMBG <sup>g</sup> | | Х | X | Х | X | Х | X | Х | X | X | Х | Х | Х | |
| 12-lead ECG <sup>h</sup> | Х | | | | | | | | Х | | | | Х | |
| Laboratory testing <sup>i</sup> | | | | | | | | | | | | | | |
| Hepatitis serology | Х | | | | | | | | | | | | | |
| FPG | Х | | Х | | Х | | Х | X | Х | X | Х | Х | Х | |

| | Screening | Period | ıble-Bl | lind Core Treatment Period <sup>a</sup> | | | | | | uble-B | Follow-up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Run-In | | | | | | | | | F | eriod <sup>b</sup> | | |
| VISIT | 1 | 2 | 3<br>Baseline | 4<br><b>2</b> | 5 | 6 <sup>€</sup> | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14<br><b>22</b> |
| Week | -4 | -2 | 0 | 1 | 4 | 8 | 12 | 18 | 26 | 39 | 52 | 65 | 79 | 81 |
| Day (window [days]) | | -14<br>(±3) | 1<br>(-) | 7<br>(±3) | 28<br>(±3) | 56<br>(±3) | 84<br>(±3) | 126<br>(±3) | 182<br>(±3) | 273<br>(±7) | 364<br>(±7) | 455<br>(±7) | 551<br>(-3 to +4) | 565<br>(±3) |
| HbA1c | Х | | Х | | X | | Х | | Х | Х | Х | Х | X | |
| Clinical chemistry, hematology <sup>j</sup> | Х | | Х | | | | Х | | Х | Х | Х | Х | Х | |
| Fasting lipids | Х | | | | | | | | X | | X | | Х | |
| Pregnancy test (WOCBP) <sup>k</sup> | Х | | Х | | X | | Х | Х | Х | Х | Х | Х | Х | |
| FSH and/or estradiol as needed <sup>k</sup> | Х | | | | | | | | | | | | | |
| Plasma concentration / | | | | | Х | | | Х | Х | | Х | | Х | |
| Urinalysis (dipstick and microscopy) <sup>m</sup> | Х | | Х | | | | | | Х | | | | Х | |
| Evaluate for glycemic rescue | | | | | | To be as | ssessed a | nd reporte | ed through | out the tr | eatment p | period | | |
| Hypoglycemia | | | | | To be asse | essed and | reported | througho | ut the stud | ły | | | | |
| AEs/SAEs/AESIs/EOSIs | | | | | To be asse | essed and | reported t | throughou | t the stud | y <mark>p</mark> | | | | |

a If a patient discontinues treatment IMP early during the 26-Week Core Treatment Period, the patient will have a Premature End-of-Treatment (EOT) Visit and a Follow-up Visit 2 weeks after the last dose of IMP. In addition, every effort will be made to have all patients return to the site at the time corresponding to their scheduled visits, particularly the Week 26 Visit. If the patient does not agree to a site visit, they will be contacted by telephone to inquire about safety status. If a patient discontinues (or completes) treatment and study at the same time, a single visit will be performed using the procedure normally planned for the EOT visit.

- b If a patient completes the Core Treatment, but discontinues IMP during the Extension Period, the patient will have a Premature EOT Visit, and a Follow-up Visit 2 weeks after the last dose of IMP. Every effort will be made to have all patients return to the site at the time corresponding to their quarterly visits (ie, every 13 weeks) during the Extension Period. At the time corresponding to their Week 79 Visit, all attempts will be made to contact the patient to inquire about safety status. If a patient discontinues (or completes) treatment and study at the same time, a single visit will be performed using the procedure normally planned for the EOT visit.
- c At Visits 4 (Week 1), 6 (Week 8) and 14 (2 weeks after the last dose of IMP) patients will be contacted by telephone, and not seen on-site.
- d Height to be measured only at screening.
- e Vital sign measurements (sitting blood pressure and heart rate): 3 separate seated blood pressure and heart rate measurements should be taken with at least 1 minute between readings, following a 5-minute rest period and prior to phlebotomy.
- f The abbreviated physical exam should focus on cardiac and respiratory systems, as well as any areas important for assessment of adverse events if necessary.
- Glucose meters used for SMBG display results as plasma glucose concentration. Patients should measure their fasting plasma glucose at least 3 times per week (including on day of each on-site study visit). After Visit 9 (Week 26), if fasting SMBG values are <120 mg/dL, over a 2-week period, the Investigator can instruct patients to self-monitor blood glucose once a week (on day of on-site study visit for weeks with on-site study visits).</p>
- h The 12-lead ECG recordings should be obtained prior to IMP administration. The ECG will be evaluated as "normal" or "abnormal".
- i All laboratory assessments occur prior to IMP administration on the day of the visit.
- j Clinical chemistry, hematology: please see list in Table 2 in protocol.
- k Serum pregnancy testing only at screening; urine pregnancy testing subsequently. Serum pregnancy test results must be reviewed prior to the Run-In phase for all WOCBP unless there is documented history of menopause (based on documented follicle-stimulating hormone [FSH] and estradiol levels if results not documented then FSH and estradiol will be tested at Screening visit) or they are surgically sterile. Any positive urine test results must be confirmed based on serum pregnancy test. The Investigator may perform additional tests at their discretion or as required by local regulations.
- Pre-dose plasma concentration samples (ie, of sotagliflozin and sotagliflozin-3-O-glucuronide) should be drawn with the other laboratory assessments at Week 4, Week 18, Week, 26, Week 52, and Week 79. Post-dose plasma concentration samples should be drawn 1 hour 30 minutes after sotagliflozin administration at Week 26 and Week 79. The date and time of the last intake of study drug prior to visits where PK samples are taken should be recorded by the patient in the patient diary. Patients should be reminded of this at visits preceding PK time points to ensure these details are captured. In the case of premature IMP discontinuation, PK samples should not be drawn at the premature EOT visit, nor at any subsequent visits.
- m Urinalysis performed by the central laboratory includes urine dipstick and microscopy. Dipstick includes assessment of specific gravity, pH, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase. Microscopy includes detection of formed cellular elements, casts, bacteria, yeast, parasites, and crystals in centrifuged urine sediment. In the event of abnormal urinalysis findings suspicious of urinary tract infection, urine culture should be performed. Positive urine culture determination will be based upon the criteria of the reporting laboratory. Additionally, urine culture should be performed if at any point the Principal Investigator suspects the presence of a UTI.
- p All SAEs, AESIs, and EOSIs will be collected starting with signing informed consent and continue until the end of the study. All AEs that occur during treatment should be followed until study completion (or until patients leave the study) or until the event has resolved, the condition has stabilized, or the patient is lost to follow-up. All patients will have a follow-up visit 2 weeks after the last dose of IMP to collect safety information.